# STATISTICAL ANALYSIS PLAN

**PROTOCOL NO: HLAB-002** 

Human Laboratory Study of ANS-6637 for Alcohol Use Disorder Protocol Version No.: 5.0 Version Date: 04Feb2020

Study Sponsor: National Institute on Alcohol Abuse and Alcoholism

Version Number 1.0 Date: 16 March 2020

# **Table of Contents**

| 1. | ABBREVIATIONS | 12 |
|---|---|---|
| 2. | INTRODUCTION | 14 |
| 3. | PROTOCOL SUMMARY 3.1. Study Objectives | |
| 4. | DEFINITION OF ANALYSIS SETS | |
| 5. | ASSSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS 5.1. Alcohol Craving Visual Analog Scales 5.2. Alcohol Consumption Endpoints 5.2.1. Daily Quantity of Alcohol Consumption 5.2.2. Drinking Days 5.2.3. Very Heavy and Heavy Drinking Day 5.2.4. Days at Risk 5.2.5. Percentage of Subjects with No Heavy Drinking Days and Percent Subjects Abstinent from Alcohol 5.2.6. Weekly Percentage of Heavy Drinking Days and Weekly Percentar Days Abstinent 5.2.7. Weekly Mean Number of Drinks and Weekly Mean Number of Drinking Day 5.2.8. World Health Organization Drinking Risk Categorical Scale 5.3. Alcohol-Related Craving, Consequences, and Withdrawal 5.4. Mood 5.5. Sleep Quality 5.6. Cigarette Smoking Quantity-Frequency and Nicotine Use Questionnaire | |
| 6. | HYPOTHESES TO BE TESTED 6.1. Primary Efficacy Endpoint 6.2. Secondary Efficacy Endpoints | 28 |
| 7. | SAMPLE SIZE CONSIDERATIONS | 29 |
| 8. | DATA QUALITY ASSURANCE | 30 |
| 9. | STATISTICAL CONSIDERATIONS 9.1. General Considerations 9.2. Participant Accountability and Protocol Deviations 9.3. Demographics and Other Baseline Characteristics 9.4. Efficacy Analysis 9.4.1. Primary Analysis of the Primary Efficacy Endpoint 9.4.2. Confirmatory Secondary Endpoints 9.4.3. Analysis of the Secondary Efficacy Endpoints 9.4.3.1. Secondary Drinking Endpoints | 31<br>31<br>32<br>32<br>32 |

| | | 9.4.3.2. Alcohol Consequences and Craving Scales | 33 |
|---|---|---|---|
| | | 9.4.3.3. Smoking and Any Nicotine Use | |
| | | 9.4.3.4. Sleep and Mood Scales | |
| | 9.5. | Handling of Missing Data | |
| | 9.6. | Safety Analysis | 35 |
| | | 9.6.1. Adverse Events | |
| | | <ul><li>9.6.2. Clinical Laboratory and Point of Care Tests</li><li>9.6.3. Vital Signs, ECG, and Body Weight</li></ul> | |
| | | 9.6.4. CIWA-AR Scores | |
| | | 9.6.5. ACQ-SF-R Scores | |
| | 9.7. | Drug Exposure and Retention Analyses | |
| | 9.8.<br>9.9. | Blood Alcohol Content | |
| | 9.9. | Exploratory Analyses | |
| | | 9.9.2 Supplemental Exploratory Analyses | |
| 10. | VALI | DATION OF PROGRAMMING CODE | |
| 11. | REFE | RENCES | 39 |
| 12. | TABL | E, LISTING, AND FIGURE SHELLS | 41 |
| | 12.1. | Tables | 41 |
| | | 12.1.1. Subject Disposition, Participation, Compliance | |
| | | <ul><li>12.1.2. Demographic and Baseline Characteristics</li><li>12.1.3. Primary Efficacy Endpoint</li></ul> | |
| | | 12.1.4. Confirmatory Secondary Efficacy Endpoints | |
| | | 12.1.5. Secondary Efficacy Endpoints | 109 |
| | | 12.1.6. Safety Analyses | |
| | 12.2. | 12.1.7. Exploratory Analyses | |
| | 12.2. | Figures | |
| | | List of Tables | |
| Table 1: | Subjec | et Disposition - All Randomized Subjects | 42 |
| Table 2: | Expos | ure to Investigational Products Using AICure Data – mITT Subjects | 44 |
| Table 3: | Total l | thm:exposure to Investigational Products Using AICure Data-Evaluable Subjects . | 44 |
| Table 4: | Comp | liance to Investigational Products Using AICure Data – mITT Subjects | 45 |
| Table 5: | Comp | liance to Investigational Products Using AICure Data – Evaluable Subjects | 45 |
| Table 6: | AiCur | e Interventions mITT Subjects | 45 |
| Table 7: | AiCu | re Interventions – Evaluable Subjects | 45 |
| Table 8: | Summ | ary of GS-54851 Blood Levels – ANS6637 Groups (mITT Subjects) | 46 |
| Table 9: | Summ | ary of GS-54851 Blood Levels – ANS6637 Groups (Evaluable Subjects) | 46 |
| Table 10: | AiCur | e Report of ANS-6637 Versus GS-5851 Blood Levels – mITT Subjects | 47 |
| Table 11: | | e Report of ANS-6637 Versus GS-5851 Blood Levels – Evaluable Subjects | 48 |
| Statistical A | Analysis I | Plan: Protocol HLAB-002, Version 1.0 Dated: 16Mar2020 4 | |

| Table 12: | Exit Interview – mITT Subjects | 48 |
|---|---|---|
| Table 13: | Exit Interview – Evaluable Subjects | 51 |
| Table 14: | Dropouts by Treatment Group and Week – mITT Subjects | 52 |
| Table 15: | Number and Percent of Subjects Using Summary Drinking Questions after Discontinuing TLFB – mITT Subjects | _ |
| Table 16: | Demographic Characteristics - mITT Subjects | 55 |
| Table 17: | Dichotomized Demographic Characteristics – mITT Subjects | 59 |
| Table 18: | Demographic Characteristics – Evaluable Subjects | 60 |
| Table 19; | Dichotomized Demographic Characteristics – Evaluable Subjects | 60 |
| Table 20: | Screening Cue Reactivity – mITT Subjects | 61 |
| Table 21: | Screening Cue Reactivity – Evaluable Subjects | 70 |
| Table 22: | Psychiatric Baseline Characteristics – mITT Subjects | 71 |
| Table 23: | Baseline POMS – mITT Subjects. | 72 |
| Table 24: | Baseline POMS – Evaluable Subjects | 75 |
| Table 25: | Baseline PSQI – mITT Subjects | 76 |
| Table 26: | Baseline PSQI – Evaluable Subjects | 76 |
| Table 27: | Baseline Drinking-related Behavior and Characteristics – mITT Subjects | 77 |
| Table 28: | Baseline Drinking-related Behavior and Characteristics – Evaluable Subjects | 79 |
| Table 29: | Baseline Drinking by TLFB – mITT Subjects | 80 |
| Table 30: | Baseline Drinking by TLFB – Evaluable Subjects | 83 |
| Table 31: | Baseline Alcohol-Related Craving, Consequences, Withdrawal and ALDH2 – mITT Subjects | 84 |
| Table 32: | Baseline Alcohol-Related Craving, Consequences, Withdrawal and ALDH2 – Evaluab Subjects | |
| Table 33: | Baseline Other Substance Use – mITT Subjects | 87 |
| Table 34: | Baseline Other Substance Use – Evaluable Subjects | 88 |
| Table 35: | Week 2 Strength of Craving Scores – mITT Subjects | 90 |
| Table 36: | Week 2 Strength of Craving <sup>1</sup> Scores – Evaluable Subjects | 91 |
| Table 37: | ANCOVA Strength of Craving <sup>1</sup> – mITT Subjects | 92 |
| Table 38: | ANCOVA Strength of Craving – Evaluable Subjects | 93 |
| Table 39: | ANCOVA Strength of Craving (Difference Alcohol-Water) – mITT Subjects | 95 |
| Table 40: | ANCOVA Strength of Craving (Difference Alcohol-Water) – Evaluable Subjects | 96 |
| Table 41: | Drinking Makes Things Perfect Scores – mITT Subjects | 96 |

| Table 42: | Drinking Makes Things Perfect Scores – Evaluable Subjects | 98 |
|---|---|---|
| Table 43: | ANCOVA Drinking Makes Things Perfect <sup>1</sup> – mITT Subjects | 99 |
| Table 44: | ANCOVA Drinking Makes Things Perfect – Evaluable Subjects | 100 |
| Table 45: | ANCOVA Drinking Makes Things Perfect <sup>1</sup> (Difference Alcohol-Water) – mITT Sub | ojects101 |
| Table 46: | ANCOVA Drinking Makes Things Perfect (Difference Alcohol-Water) – Evaluable Subjects | 102 |
| Table 47: | Drink Now Scores- mITT Subjects | 103 |
| Table 48: | Drink Now Scores – Evaluable Subjects | 104 |
| Table 49: | ANCOVA Drink Now <sup>1</sup> – mITT Subjects | 105 |
| Table 50: | ANCOVA Drink Now <sup>1</sup> – Evaluable Subjects | 106 |
| Table 51: | ANCOVA Drink Now <sup>1</sup> (Difference Alcohol-Water) – mITT Subjects | 106 |
| Table 52: | ANCOVA Drink Now <sup>1</sup> (Difference Alcohol-Water) – Evaluable Subjects | 106 |
| Table 53: | Turn Down Drink Scores – mITT Subjects | 106 |
| Table 54: | Turn Down Drink Scores – Evaluable Subjects | 106 |
| Table 55: | ANCOVA Turn Down Drink <sup>1</sup> – mITT Subjects | 107 |
| Table 56: | ANCOVA Turn Down Drink <sup>1</sup> – Evaluable Subjects | 107 |
| Table 57: | ANCOVA Turn Down Drink <sup>1</sup> (Difference Alcohol-Water) – mITT Subjects | 107 |
| Table 58: | ANCOVA Turn Down Drink <sup>1</sup> (Difference Alcohol-Water) – Evaluable Subjects | 107 |
| Table 59: | Average of Cue Scores – mITT Subjects | 107 |
| Table 60: | Average of Cue Scores – Evaluable Subjects. | 107 |
| Table 61: | ANCOVA Average of Cue Scores <sup>1</sup> – mITT Subjects | 107 |
| Table 62: | ANCOVA Average of Cue Scores <sup>1</sup> – Evaluable Subjects | 107 |
| Table 63: | ANCOVA Average of Cue Scores <sup>1</sup> (Difference Alcohol-Water) – mITT Subjects | 107 |
| Table 64: | ANCOVA Average of Cue Scores <sup>1</sup> (Difference Alcohol-Water) – Evaluable Subjects | s 107 |
| Table 65: | Beverage Liking Scores – mITT Subjects | 108 |
| Table 66: | Beverage Liking Scores – Evaluable Subjects | 108 |
| Table 67: | Percentage of Subjects No Heavy Drinking Days Weeks 2-5 – mITT Subjects | 110 |
| Table 68: | Percentage of Subjects with No Heavy Drinking Days Weeks 2-5 – Full Model Logis Regression (mITT) | |
| Table 69: | Percentage of Subjects Abstinent from Alcohol Weeks 2-5 – mITT Subjects | 111 |
| Table 70: | Percentage of Subjects Abstinent from Alcohol Weeks 2-5 – Full Model Logistic Regression (mITT) | 112 |
| Table 71: | WHO 1-Level Decrease in Alcohol Consumption (mITT) – Weeks 2-5 | 112 |

| Table 72: | WHO 1-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 2-5 | 113 |
|---|---|---|
| Table 73: | WHO 2-Level Decrease in Alcohol Consumption (mITT) – Weeks 2-5 | 114 |
| Table 74: | WHO 2-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 2-5 | 114 |
| Table 75: | Percentage of Days Abstinent per Week (mITT) – Weeks 2-5 | 114 |
| Table 76: | Percentage of Days Abstinent per Week (mITT) Full Model, Mixed Effects, Weeks | 2-5115 |
| Table 77: | Percentage of Heavy Drinking Days per Week (mITT) – Weeks 2-5 | 118 |
| Table 78: | Percentage of Heavy Drinking Days per Week (mITT) – Full Model, Mixed Effects, Weeks 2-5 | 118 |
| Table 79: | Percentage of Very Heavy Drinking Days per Week (mITT) – Weeks 2-5 | 118 |
| Table 80: | Percentage of Very Heavy Drinking Days per Week (mITT) – Full Model, Mixed Eff<br>Weeks 2-5 | |
| Table 81: | Drinks per Week (mITT) – Weeks 2-5. | 118 |
| Table 82: | Drinks per Week (mITT) – Full Model, Mixed Effects, Weeks 2-5 | 118 |
| Table 83: | Drinks per Drinking Day (mITT) – Weeks 2-5 | 118 |
| Table 84: | Drinks per Drinking Day (mITT) – Full Model, Mixed Effects, Weeks 2-5 | 118 |
| Table 85: | Mean Cigarettes Smoked Among Smokers (mITT) – Weeks 2-5 | 118 |
| Table 86: | Mean Cigarettes Smoked Among Smokers (mITT) – Full Model, Mixed Effects, Wee 5 | |
| Table 87: | PACS (mITT) – Weeks 2-5 | 118 |
| Table 88: | PACS (mITT) – Full Model, Mixed Effects, Weeks 2-5 | 118 |
| Table 89: | Percentage of Subjects Abstinent from Nicotine Use <sup>1</sup> Weeks 2-5 – Among Subjects the Used Nicotine Products at Baseline | |
| Table 90: | Percentage of Subjects Abstinent from Nicotine Use <sup>1</sup> Weeks 2-5 – Full Model Logisti Regression (Among Nicotine Users at Baseline) | |
| Table 91: | Percentage of Subjects Abstinent from Smoking Weeks 2-5 – Among Baseline Smoke | ers121 |
| Table 92: | Percentage of Subjects Abstinent from Smoking Weeks 2-5 – Full Model Logistic Regression (Among Baseline Smokers) | 121 |
| Table 93: | PSQI Scores – mITT Subjects | 121 |
| Table 94: | ANCOVA PSQI Score – mITT Subjects | 121 |
| Table 95: | POMS Total Mood Disturbance Score – mITT. | 123 |
| Table 96: | POMS Total Mood Disturbance Score (mITT) – Full Model, Mixed Effects, Weeks 4 | + 6123 |
| Table 97: | POMS Tension-Anxiety Score – mITT Subjects | 126 |
| Table 98:<br>Statistical A | POMS Tension-Anxiety Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6 Analysis Plan: Protocol HLAB-002, Version 1.0 Dated: 16Mar2020 7 | 126 |

| Table 99: | POMS Anger-Hostility Score – mITT Subjects |
|---|---|
| Table 100: | POMS Anger-Hostility Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6 126 |
| Table 101: | POMS Vigor-Activity Score – mITT Subjects |
| Table 102: | POMS Vigor-Activity Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6 126 |
| Table 103: | POMS Fatigue-Inertia Score – mITT Subjects |
| Table 104: | POMS Fatigue-Inertia Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6 126 |
| Table 105 | POMS Confusion-Bewilderment Score – mITT Subjects |
| Table 106: | POMS Confusion-Bewilderment Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6126 |
| Table 107: | POMS Depression-Dejection Score – mITT Subjects |
| Table 108: | POMS Depression-Dejection Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6.126 |
| Table 109: | PROMIS Negative Consequences of Alcohol Scores – mITT Subjects |
| Table 110: | ANCOVA PROMIS Negative Consequences of Alcohol – mITT Subjects |
| Table 111: | Overall Summary of Adverse Events – Safety Subjects |
| Table 112: | Overall Summary of Adverse Events p-values – Safety Subjects |
| Table 113: | Number and Percentage of Subjects with Adverse Events - Safety Subjects |
| Table 114: | Number and Percentage of Subjects with Adverse Events p-values - Safety Subjects 132 |
| Table 115: | Number and Percentage of Subjects with Adverse Events by ALDH2 Status – Safety Subjects |
| Table 116: | Number and Percentage of Subjects with Adverse Events by Treatment Arm - ALDH2 Deficient Subjects |
| Table 117: | Number and Percentage of Subjects with Adverse Events by Treatment Arm p-values - ALDH2 Deficient Subjects |
| Table 118: | Number and Percentage of Subjects with Adverse Events by Treatment Arm - ALDH2 Non-Deficient Subjects |
| Table 119: | Number and Percentage of Subjects with Adverse Events by Treatment Arm p-values - ALDH2 Non-Deficient Subjects |
| Table 120: | Number and Percentage of Subjects Taking Drugs with Potential for Interaction |
| Table 121: | Elicited Adverse Event Questions – Safety Subjects |
| Table 122: | Elicited Adverse Event Questions p-values – Safety Subjects |
| Table 123: | Number of Elicited Adverse Events – Safety Subjects |
| Table 124: | Summary of Subjects with Adverse Events by Severity and Relationship – Placebo 137 |
| Table 125: | Summary of Subjects with Adverse Events by Severity and Relationship – ANS-6637 200 mg |

| Table 126: | Summary of Subjects with Adverse Events by Severity and Relationship – ANS-6637 600 mg |
|---|---|
| Table 127: | Number and Percentage of Subjects with Adverse Events by Maximum Severity - Safety Subjects |
| Table 128: | Number and Percentage of Subjects Adverse Events by Relatedness - Safety Subjects 140 |
| Table 129: | Number and Percentage of Subjects with Treatment-Related Adverse Events by Maximum Severity- Safety Subjects |
| Table 130: | Number and Percentage of Subjects with Adverse Events Occurring in >= 10% of Subjects in Any One Group - Safety Subjects |
| Table 131: | Number and Percentage of Subjects with Adverse Events Occurring in >= 10% of Subjects in Any One Group p-values - Safety Subjects |
| Table 132: | Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study - Safety Subjects |
| Table 133: | Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study Medication – Safety Subjects |
| Table 134: | CIWA-AR Score > 10 at Least Once During Treatment – Safety Subjects |
| Table 135: | Summary of Vital Signs and Body Weights – Safety Subjects |
| Table 136: | Summary of ECG Results - Safety Subjects |
| Table 137: | Summary of Blood Chemistries and Thyroid Function – Safety Subjects |
| Table 138: | Summary of Urinalysis Continuous Data – Safety Subjects |
| Table 139: | Summary of Urine Glucose and Nitrites – Safety Subjects |
| Table 140: | Summary of Urine Protein, Ketones, Billirubin, Leukocyte Esterace, and Blood – Safety Subjects |
| Table 141: | Summary of Positive Urine Drug Tests, Preganancy Test or BAC > 0.02 Any Time During the Study– Safety Subjects |
| Table 142: | Frequency of Subjects with Suicidal Ideation Any Time During the Study – Safety Subjects |
| Table 143: | Return to Baseline ACQ-SF-R Scores – Safety Subjects |
| Table 144: | Difference Between First and Second Alcohol Cues – mITT Subjects |
| | List of Listings |
| Listing 1: Su | bject Disposition - All Subjects |
| Listing 2. Er | arollment and Randomization – All Consented Subjects |

| Listing 3: Reason not Eligible – Screen Failures | 159 |
|---|---|
| Listing 4: Protocol Deviations – Safety Subjects | 160 |
| Listing 5: Subjects Excluded from the Efficacy Analysis or Evaluable Set | 161 |
| Listing 6: Demographics Data – Safety Subjects | 162 |
| Listing 7: Baseline Drinking Characteristics – mITT Subjects | 164 |
| Listing 8: Baseline Smoking Characteristics – mITT Subjects | 166 |
| Listing 9: MINI DSM5 Disorders – Safety Subjects | 166 |
| Listing 10: MINI DSM-5 AUD – Safety Subjects | 167 |
| Listing 11: Medical History – Safety Subjects | 167 |
| Listing 12: Drinking Goal – mITT Subjects | 168 |
| Listing 13: Physical Exam – Safety Subjects | 168 |
| Listing 14: Daily and Weekly Standard Drink Units (TLFB) During Treatment – mITT Subjects | 169 |
| Listing 15: Brief Drinking Questionnaire – mITT Subjects | 169 |
| Listing 16: Cue Reactivity – mITT Subjects | 170 |
| Listing 17: Cue Session Beverage – mITT Subjects | 171 |
| Listing 18: Drinking Consequences and Craving Scores – mITT Subjects | 172 |
| Listing 19: Pittsburg Sleep Quality Index Scores – mITT Subjects | 172 |
| Listing 20: Smoking and Other Nicotine Use Data- mITT Subjects | 173 |
| Listing 21: MINI AUD- Safety Subjects | 174 |
| Listing 22. Exit Interview – mITT Subjects | 175 |
| Listing 23: Drug Exposure from AiCure- mITT Subjects. | 177 |
| Listing 24: Drug Accountability – Safety Subjects | 177 |
| Listing 25: Take Control – mITT Subjects | 178 |
| Listing 26: Adverse Events – Safety Subjects | 179 |
| Listing 27: Adverse Events – Subjects Taking CYP3A Substrate | 180 |
| Listing 28: Serious Adverse Events – Safety Subjects | 181 |
| Listing 29: Elicited Adverse Events – Safety Subjects | 183 |
| Listing 30: POMS Scores – mITT Subjects | 183 |
| Listing 31. Columbia-Suicide Severity Scale – Safety Subjects | 184 |
| Listing 32: Blood Chemistries and Thyroid Results – Safety Subjects | 186 |
| Listing 33: Hematology – Safety Subjects | 187 |
| Listing 35: Urinalysis – Safety Subjects | 188 |

| Listing 35: 1 | Jrinalysis Microscopy <sup>1</sup> – Safety Subjects | 189 |
|---|---|---|
| Listing 36: 1 | Pregnancy Test/Birth Control Data – Safety Subjects | 190 |
| Listing 37: 1 | Blood Alcohol Concentration – Safety Subjects | 191 |
| Listing 38. U | Jrine Drug Screen – Safety Subjects | 191 |
| Listing 39: \ | Vital Signs and Body Weights- Safety Subjects | 192 |
| Listing 40. I | ECG – Safety Subjects | 193 |
| Listing 41. I | Prior and Concomitant Medications – Safety Subjects | 194 |
| Listing 42: 1 | Blood for Drug Concentrations – Safety Subjects | 194 |
| Listing 43: | Comments – Safety Subjects | 195 |
| | List of Figures | |
| Figure 1: | Percentage of Subjects No Heavy Drinking Days Weeks 2-5 | 197 |
| Figure 2: | Percentage of Subjects Abstinent Weeks 2-5 | 197 |
| Figure 3: | Weekly Percentage of Subjects No Heavy Drinking Days (mITT) | 197 |
| Figure 4: | Weekly Percentage of Subjects Abstinent (mITT) | 197 |
| Figure 5: | Weekly Percentage WHO 1-Level Decrease in Alcohol Consumption (mITT) | 197 |
| Figure 6: | Weekly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT) | 197 |
| Figure 7: | Percentage Days Abstinent per Week Least Squares Means – (mITT) | 197 |
| Figure 8: | Percent Heavy Drinking Days per Week Lease Squares Means –(mITT) | 197 |
| Figure 9: | Mean Drinks per Week Lease Squares Means – (mITT) | 197 |
| Figure 10: | Mean Drinks per Drinking Day by Week Least Squares Means – (mITT) | 197 |
| Figure 11: | Weekly Number of Cigarettes Smoked in Smokers Over Entire Treatment Period – L<br>Squares Means (mITT) | |
| Figure 12: | Clinical Chemistry, Urinalysis, and Hematology Values Over Time | 197 |

# 1. ABBREVIATIONS

| Abbreviation | Definition | |
|---|---|---|
| ACQ-SF-R | Alcohol Craving Scale – Short Form | |
| AE | Adverse event | |
| AICc | Akaike Information Criterion corrected for finite samples | |
| ALDH2 | Aldehyde dehydrogenase 2 | |
| ALT | Alanine aminotransferase | |
| ANOVA | Analysis of variance | |
| ANCOVA | Analysis of covariance | |
| AST | Aspartate aminotransferase | |
| AUD | Alcohol Use Disorder | |
| BAC | Blood alcohol concentration | |
| CI | Confidence interval | |
| CIWA-AR | Clinical Institute Withdrawal Assessment for Alcohol-revised | |
| CrCl | Creatinine clearance | |
| C-SSRS | Columbia-Suicide Severity Rating Scale | |
| CTCAE | Common terminology criteria for adverse events | |
| dL | Deciliter | |
| DSM-5 | Diagnostic and Statistical Manual of Mental Disorders – Fifth Edition | |
| ECG | Electrocardiogram | |
| eCRF | Electronic Case Report Form | |
| EDMS | Electronic Data Management System | |
| EOS | End of study | |
| F | Fahrenheit | |
| FDA | Food and Drug Administration | |
| g | Gram | |
| GGT | Gamma-glutamyl transferase | |
| hr | Hour | |
| ICH | International Conference on Harmonization | |
| MedDRA | Medical Dictionary for Regulatory Activities | |
| mg | Milligram | |
| μg | Microgram | |
| min | Minutes | |
| MINI | MINI Neuropsychiatric Interview | |
| mITT | Modified intention-to-treat | |
| mL | Milliliter | |
| mm | Millimeter | |
| NHDD | No heavy drinking days | |
| NIAAA | National Institutes on Alcohol Abuse and Alcoholism | |
| OZ | Ounce | |
| Statistical Analy | rsis Plan: Protocol HLAB-002. Version 1.0 Dated: 16Mar2020 | 12 |

| Abbreviation | Definition |
|--------------|----------------------------------------------------------|
| PACS | Penn Alcohol Craving Scale |
| POMS | Profile of Mood State |
| PROMIS | Patient Reported Outcomes Measurement Information System |
| PSNHDD | Percentage of subjects with no heavy drinking days |
| PSQI | Pittsburg Sleep Quality Index |
| PT | Preferred term |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SDU | Standard drinking unit |
| SOC | System Organ Class |
| THC | Tetrahydrocannabinol |
| TLFB | Timeline followback |
| TSH | Thyroid-stimulating hormone |
| ULN | Upper limit of normal |
| VAS | Visual analog scale |
| WHO | World Health Organization |

#### 2. INTRODUCTION

This statistical analysis plan (SAP) for Protocol No. HLAB-002, "Human Laboratory Study of ANS-6637 for Alcohol Use Disorder" describes and expands upon the analytical plan presented in the protocol.

This document contains all planned analyses, reasons and justifications for these analyses for all study data. This plan also includes sample tables, figures, and listings that will be populated. The SAP will follow the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines as indicated in Topic E3 (Structure and Content of Clinical Study Reports), Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH.

The following sources were used in preparation of this SAP:

- Protocol # HLAB-002, Protocol Version No.: 5.0; Version Date: 04 Feb 2020
- ICH Guidance Topics E9, E3 and E8

#### 3. PROTOCOL SUMMARY

## 3.1. Study Objectives

# **3.1.1. Primary**

The primary objective of this study is to evaluate the effects of two different doses of ANS-6637, 200 mg (given as 2 x 100 mg tablet) and 600 mg (given as 2 x 300 mg tablet) once a day, and matched placebo, on alcohol cue-elicited alcohol craving during a human laboratory paradigm after 1 week of daily dosing among subjects with moderate to severe alcohol use disorder (AUD) as confirmed by the Diagnostic and Statistical Manual of Mental Disorders – Fifth Edition (DSM-5<sup>TM</sup>).

## 3.1.2. Secondary

Secondary objectives include evaluation of ANS-6637 200 mg once-daily, ANS-6637 600 mg once daily, and matched placebo on reduction of alcohol consumption, alcohol craving weekly (PACS), cigarette smoking (among smokers), nicotine use (among nicotine users), mood, sleep, study retention, alcohol negative consequences, and safety and tolerability throughout the last 4 weeks of the treatment period.

## 3.2. Study Design

This study is a 3-arm, double-blind, randomized, placebo-controlled, parallel group, 3-site study designed to assess the effects of ANS-6637 as compared with placebo on responses to in vivo alcohol cue exposure in the human laboratory setting. After signing informed consent, subjects will be screened for eligibility and have other baseline assessments. Screening is permitted over a 14-day period and most baseline assessments will be performed on the day of randomization. Assessments include alcohol breathalyzer test (before signing consent), medical history, physical examination, vital signs, electrocardiogram (ECG), drinking history by the timeline follow-back (TLFB) method, Clinical Institute Withdrawal Assessment for Alcohol-revised (CIWA-AR), prior medication use, MINI neuropsychiatric interview, urine drug test, smoking quantity frequency and nicotine use interview, clinical laboratory tests including chemistry, hematology, thyroid function tests, and medical urinalysis, craving responses during cue reactivity session, Columbia Suicide Severity Rating Scale (C-SSRS), drinking goal, Penn Alcohol Craving Scale (PACS), Pittsburg Sleep Quality Index (PSQI), PROMIS Alcohol Negative Consequences short form, Profile of Moods State (POMS), blood sample for aldehyde dehydrogenase 2 (ALDH2) deficiency genetic test and confirmation that subjects are treatment seeking and desire a reduction or cessation of drinking. Women of child-bearing potential will have a pregnancy test.

If eligible for the study, 81 subjects will be randomized using a stratified permuted block randomization procedure in an approximate 1:1:1 ratio (targeting 27 subjects per group and 27 subjects per each of 3 clinical sites) to receive either ANS-6637 200 mg once daily, ANS-6637 600 mg once daily, or matched placebo for 5 weeks. Subjects will be seen in the clinic at screening, at randomization and 5 other times during the study. A final follow-up telephone interview will occur 2 weeks after the end of study in-clinic visit.

| Study assessments and procedures will be performed at the visits and time points outlined in the Schedule of Assessments ( <b>Table 1</b> ). |
|---|

**Table 1:** Schedule of Assessments

| Study Phase | Screening | Treatment | | | | | End of Study <sup>a</sup> | Follow-up<br>Call |
|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 1 | 2 | 3 | 4 | 5 | 6 | 7 | |
| Study Week (Days) <sup>b</sup> | -2 to -1<br>(-14 to -1) | 1<br>(1 to 7) | 2<br>(8 to 14) | 3<br>(15 to 21) | 4<br>(22 to 28) | 5<br>(29 to 35) | 6<br>(36 to 42) | 8<br>(50 to 56) |
| Informed Consent | X | | | | | | | |
| Alcohol Breathalyzer | X | X | X | X | X | X | X | |
| Urine Drug Test <sup>c</sup> | X | X | X | X | X | X | X | |
| Locator Form | X | Update | Update | Update | Update | Update | Update | |
| Demographics | X | | | | | | | |
| Medical History | X | Update | | | | | | |
| Physical Exam | X | Update | | | | | | |
| Body Weight | X | X | X | X | X | X | X | |
| MINI V 7.0 | X | | | | | | | |
| C-SSRS | | X | X | X | X | X | X | |
| Clinical Chemistry <sup>d</sup> | X | | X | X | X | X | X | |
| Hematology <sup>e</sup> | X | | | X | | | X | |
| Thyroid Function Tests <sup>f</sup> | X | | X | X | X | X | X | |
| Medical Urinalysis | X | | | X | | | X | |
| Pregnancy Test | X | X | X | X | X | X | X | |
| Birth control methods (all subjects) | X | X | X | X | X | X | X | |
| Vital Signs <sup>g</sup> | X | X | X | X | X | X | X | |
| Eligibility Checklist | X | X | | | | | | |
| Drinking Goal | | X | | | | | | |
| ECG | X | | | X | | | X | |
| Prior and Concomitant Meds | X | X | X | X | X | X | X | X |

Statistical Analysis Plan: Protocol HLAB-002, Version 1.0 Dated: 16Mar2020

| Study Phase | Screening | Treatment | | | | | End of Study <sup>a</sup> | Follow-up<br>Call |
|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | 1 | 2 | 3 | 4 | 5 | 6 | 7 | |
| Study Week (Days) <sup>b</sup> | -2 to -1<br>(-14 to -1) | 1<br>(1 to 7) | 2<br>(8 to 14) | 3<br>(15 to 21) | 4<br>(22 to 28) | 5<br>(29 to 35) | 6<br>(36 to 42) | 8<br>(50 to 56) |
| CIWA-AR | X | X | X | X | X | X | X | X |
| Screening Cue Reactivity Session:<br>VAS Scales, typical alcoholic<br>beverage | X | | | | | | | |
| Pharmacogenetic sampling (ALDH2) | | X | | | | | | |
| Randomization | | X (Day 1) | | | | | | |
| Blood for Drug Concentration | | | X | | X | | | |
| Drug compliance/ accountability/<br>Review AiCure | | Dispense<br>Day 1 | X | X | X | X | X | |
| AEs (open ended question) and elicited AE questions | | X | X | X | X | X | X | X |
| Brief Telephone Interview <sup>h</sup> | | 2 times<br>during the<br>week | As needed if the subject misses a clinic visit | | | | | |
| Take Control | | X | X | X <sup>i</sup> | X | X | X | |
| Treatment Cue Reactivity Session:<br>VAS Scales, typical alcoholic<br>beverage | | | X | | | | | |
| TLFB | X | X | X | X | X | X | X | |
| Brief Drinking Questionnaire | AS NEEDED | | | | | | | |
| Exit Interview | | | | | | | X | |
| ACQ-SF-R | 2X pre/post<br>cue session | | 2X<br>pre/post<br>cue<br>session | | | | | |
| PACS | | X | X | X | X | X | X | |

| Study Phase | Screening 1 | Treatment | | | | | End of Study <sup>a</sup> | Follow-up<br>Call |
|---|---|---|---|---|---|---|---|---|
| Clinic Visit # | | 2 | 3 | 4 | 5 | 6 | 7 | |
| Study Week (Days) <sup>b</sup> | -2 to -1<br>(-14 to -1) | 1<br>(1 to 7) | 2<br>(8 to 14) | 3<br>(15 to 21) | 4<br>(22 to 28) | 5<br>(29 to 35) | 6<br>(36 to 42) | 8<br>(50 to 56) |
| Smoking quantity/frequency and nicotine use | | X | X | X | X | X | X | |
| PSQI | | X | | | | | X | |
| POMS | | X | | | X | | X | |
| PROMIS Alcohol Negative<br>Consequences | | X | | | | | X | |
| Treatment Referral | | | | | | | X | |
| Follow-Up Telephone Interview | | | | | | | | X |
| Final Subject Disposition | | | | | | | | X |

<sup>&</sup>lt;sup>a</sup> EOS - end of study. These assessments are to be done at Week 6 or if the subject discontinues early and agrees to a final clinic visit.

<sup>&</sup>lt;sup>b</sup> Within each study week, there should be a least two days elapsed since the visit in the prior week.

<sup>&</sup>lt;sup>c</sup> Test for opiates (i.e., morphine test), cocaine, amphetamines, methamphetamine, THC, buprenorphine, methadone, benzodiazepines, oxycodone, barbiturates, 3,4-methylenedioxy-methamphetamine (MDMA – also known as ecstasy), and EtG.

d AST, ALT, alkaline phosphatase, total bilirubin, creatinine, gamma glutamyl transferase (GGT), and albumin. CrCl will also be calculated each time creatine is measured.

<sup>&</sup>lt;sup>e</sup> Hematology tests include complete blood cell count with differential.

f The thyroid panel includes: thyroid-stimulating hormone (TSH), thyroxine (T4) and free thyroxine (free T4), and triiodothyronine (T3).

<sup>&</sup>lt;sup>g</sup> Sitting blood pressure and heart rate.

h AEs, concomitant medications, CIWA-AR, and drug compliance reminder. Telephone calls during the first week, should be separated by at least one day between calls, and will include assessments for AEs, concomitant medications, CIWA-AR, and a drug compliance reminder. The second call should be several days before the cue session to remind the subject of the planned visit.

<sup>&</sup>lt;sup>1</sup> Two Take Control modules will be viewed at this visit.

#### 3.3. Study Endpoints

## 3.3.1. Primary Efficacy Endpoint

The primary efficacy endpoint is the "strength" of alcohol craving VAS score (item 1 below) upon presentation of the first alcohol cue at Week 2 – after one week of investigational product treatment.

Confirmatory secondary endpoints include the VAS score for the other 3 VAS scales (items 2 through 4 below) for the first alcohol cue and the average score of the 4 VAS craving items; and the difference score (alcohol craving VAS scores minus the water craving VAS score). The also a confirmatory secondary endpoint. The 4 VAS craving items in the order of presentation are:

- 1. How strong is your craving to drink alcohol? note this is the primary efficacy endpoint.
- 2. Having a drink would make things just perfect.
- 3. If I could drink alcohol now, I would drink it.
- 4. It would be hard to turn down a drink right now.

The beverage liking item is: How much did you like the beverage just given to you?

## 3.3.2. Secondary Efficacy Endpoints

Secondary efficacy endpoints will be analyzed over the last 4 weeks of the treatment period of treatment.

- 1. Percentage of subjects with no heavy drinking days. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
- 2. Percentage of subjects abstinent from alcohol
- 3. Percentage of subjects with at least a WHO 2-level decrease in alcohol consumption
- 4. Percentage of subjects with at least a WHO 1-level decrease in alcohol consumption
- 5. Percentage of days abstinent per week
- 6. Percentage of heavy drinking days per week
- 7. Percentage of very heavy drinking days per week. A "very heavy drinking day" is 8 or more drinks per drinking day for women and 10 or more drinks per drinking day for men.
- 8. Weekly mean number of drinks per week
- 9. Weekly mean drinks per drinking day
- 10. Cigarettes smoked per week among smokers
- 11. Percentage of subjects with no nicotine use among those reporting nicotine use at baseline
- 12. Alcohol craving score (PACS)
- 13. Sleep quality (PSQI) score

- 14. Profile of Mood States (POMS) score
- 15. PROMIS Alcohol Negative Consequences Score

#### 3.3.3. Safety Endpoints

- 1. Vital signs
- 2. Body weight
- 3. Clinical laboratory parameters
- 4. BAC by breathalyzer
- 5. Urine drug tests
- 6. AEs and elicited AEs (flushing or heat sensation, heart rate increases or heart palpitations, and appetite change and AEs in subjects taking CYP3A-sensitive substrates)
- 7. ECG results
- 8. CIWA-AR scores
- 9. Frequency of subjects with suicidal ideation at any time during the treatment period (C-SSRS)
- 10. Concomitant medication use
- 11. ACQ-SF-SR score (pre- and post-cue response sessions)

## 3.3.4. Compliance

Compliance will be assessed using the AiCure smart phone application and by tablet counts of returned bottles at regular clinic visits. In addition, blood will be collected to determine plasma levels of GS-548351. Compliance will be calculated as the percentage of investigational products taken as prescribed and by the total amount of medication consumed. Participation in study visits will be evaluated as the percentage of subjects with complete drinking data. Compliance determined by GS-548351 plasma levels will be reported as number and percentage of subjects with a level above the limit of detection at each time point.

#### 4. **DEFINITION OF ANALYSIS SETS**

The study analysis populations will consist of the following:

**Modified Intention-to-Treat (mITT) Analysis Set:** The mITT set is defined as subjects randomized to participate in the study that took at least one dose of investigational product and had a non-missing VAS craving primary endpoint.

**Evaluable Analysis Set:** The evaluable analysis set for the secondary endpoints is defined as those subjects randomized to the study who took at least 2 tablets per day for at least 80% of days in Weeks 1-5.

**Safety Analysis Set:** The safety analysis set includes all subjects who took at least one dose of investigational product.

The analysis of the primary and confirmatory efficacy endpoints will be conducted on both the mITT and evaluable analysis sets. Secondary endpoint analyses will be performed on the mITT set only. Safety analyses will be conducted on the safety analysis set.

#### 5. ASSSESSMENT AND JUSTIFICATION OF STUDY ENDPOINTS

#### **5.1.** Alcohol Craving Visual Analog Scales

Alcohol craving in response to a water and typical alcohol beverage cue is assessed using 4 individual VAS items adapted from the ACQ (Singleton-1994).

The VAS craving scale items include in the following order:

- 1. How strong is your craving to drink alcohol?
- 2. Having a drink would make things just perfect.
- 3. If I could drink alcohol now, I would drink it.
- 4. It would be hard to turn down a drink right now.

Anchors (scores) for items 1, 3, and 4 are: Strongly Disagree (0) to Strongly Agree (20).

Anchors (scores) for question 2 are: None (0) to Extremely Strong (20).

Since the typical alcohol beverage is presented twice, the first presentation and associated VAS is to be used in the analysis.

There will be no imputation for missing values.

# **5.2.** Alcohol Consumption Endpoints

### 5.2.1. Daily Quantity of Alcohol Consumption

Drinking will be assessed using the TLFB methodology and Form 90 structured assessment pattern chart. The TLFB is a semi-structured interview that provides estimates of the daily quantity of alcohol consumption during specified time periods. It uses a calendar prompt and a number of other memory aids (e.g., holidays, payday, and other personally relevant dates) to facilitate accurate recall of drinking or other drug use during the target period. The procedure has been widely used in clinical and research contexts. It has demonstrated adequate levels of reliability and validity when administered as an in-person interview, over the telephone, and when administered via computer (Carey-1997, Sobell et al-1988, Sobell et al-1996).

If a subject is withdrawn from the study early and is no longer participating in clinic visits or providing TLFB drinking data but is willing to be contacted by phone at the week most proximal to dropout, then they will be asked about any drinking and heavy drinking during the time since last contact. Phone calls will continue until the end of the treatment period, as deemed acceptable by the patient. The two questions cover whether the subject had any heavy drinking days or drinking days during the period covered and will be used to capture drinking data in the absence of individual daily TLFB drinking data.

#### 5.2.2. Drinking Days

A drinking day is one calendar day in which the subject reported any alcohol consumption (i.e., > 0 standard drinking units [SDUs]). A standard drink contains approximately 0.6 fluid ounces (oz) of pure alcohol. The data given by the subjects on amount and type of alcoholic beverage(s) consumed will be converted to SDUs. Standard drink unit definitions are provided in **Table 2**. Statistical Analysis Plan: Protocol HLAB-002, Version 1.0 Dated: 16Mar2020

#### **Table 2:** Standard Drink Unit Definitions

For Beer ( $\sim 5\%$  alcohol), the approximate number of SDUs in:

- 12 oz = 1.0
- 16 oz = 1.3
- 24 oz = 2.0
- 40 oz = 3.3

For malt liquor (~ 7% alcohol), the approximate number of SDUs in:

- 12 oz = 1.4
- 16 oz = 1.9
- 22 oz = 2.6
- 40 oz = 4.7

For table wine (~ 12% alcohol), the approximate number of SDUs in:

- 750 mL bottle = 250z = 5.0
- 5 oz glass = 1.0
- 10 oz glass = 2.0

For 80 proof spirits (~ 40% alcohol), or hard liquor, the approximate number of SDUs in:

- 1.5 oz (mixed drink) = 1.0
- 16 oz (pint) = 8.5
- 25 oz (a fifth) = 17.0
- 1.75 L (59 oz) = 39.0

#### 5.2.3. Very Heavy and Heavy Drinking Day

A very heavy drinking day is defined as 8 or more drinks per day for a woman, and 10 or more for men. A heavy drinking day is defined as a day with 5 or more drinks (SDUs) for males and 4 or more drinks (SDUs) for females.

#### 5.2.4. Days at Risk

If a subject is being treated at an inpatient facility, is incarcerated, or otherwise under confinement, the days spent in under these conditions is considered a reduction in the days at risk for drinking and is deducted from the denominator in calculations of rates of drinking days.

# 5.2.5. Percentage of Subjects with No Heavy Drinking Days and Percentage of Subjects Abstinent from Alcohol

The percentage of subjects with no heavy drinking days is the number of subjects that have no heavy drinking days during the period of interest divided by the number of subjects with at least one day of non-missing drinking data during the period of interest, multiplied by 100.

The percentage of subjects abstinent from alcohol is calculated similarly, except the numerator is the number of subjects that have no drinking days during the period of interest.

# 5.2.6. Weekly Percentage of Heavy Drinking Days and Weekly Percentage of Days Abstinent

Weekly percentage of heavy drinking days is the number of heavy drinking days in a 7-day period divided by 7 then multiplied by 100. The TLFB permits capturing data in a subsequent visit if a visit is missed; however, if fewer than 7 days are observed then the denominator is the number of days observed in the 7-day period. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly percentage of days abstinent is similarly calculated by using the number of days abstinent instead of the number of heavy drinking days.

# 5.2.7. Weekly Mean Number of Drinks and Weekly Mean Number of Drinks per Drinking Day

Weekly mean number of drinks is the sum of SDUs calculated to the tenths over 7 calendar days divided by the number of days with non-missing data. The quotient is multiplied by 7. At least 3 days in a week must be observed; otherwise, the week is considered missing.

Weekly mean number of drinks per drinking days utilizes the same numerator, and the denominator is the number of days with greater than 0 SDUs. Weeks where all days within the week are abstinent are assigned a value of 0 for weekly drinks per drinking day.

# 5.2.8. World Health Organization Drinking Risk Categorical Scale

The WHO has developed a drinking risk categorical scale that can be used in a responder analysis approach to assess clinically relevant decreases in alcohol consumption (<u>Aubin et al-2015</u>). Two dichotomous endpoints will be analyzed: WHO 1-level and WHO 2-level decrease in alcohol consumption. The WHO 1-level and 2-level decrease endpoints are the percentage of subjects experiencing at least a 1-level or 2-level decrease in WHO levels of alcohol consumption, respectively, from the level at baseline (the period including the 28 days before screening) to the level during the last 4 weeks of the maintenance phase (Study Weeks 2-5). The WHO levels of average alcohol consumption per day are as follows:

| | Males | Females |
|----------------|------------|-----------|
| Low Risk | 1 to 40g | 1 to 20g |
| Medium Risk | 41 to 60g | 21 to 40g |
| High Risk | 61 to 100g | 41 to 60g |
| Very High Risk | 61+g | |

where 14g = 1 SDU (<u>WHO-2000</u>). In computing the alcohol consumption level, average drinks per day will be used, computed as the sum of all drinking in the 28 day period divided by the number of days with non-missing drinking data in that period. Abstinent subjects will be included in a separate "Abstinent" category. A subject must have at least 1 week of data during the last 4 weeks of the maintenance phase to be considered non-missing.

# 5.3. Alcohol-Related Craving, Consequences, and Withdrawal

Alcohol-related craving is measured using the ACQ-SF-R scale and PACS; alcohol-related consequences are measured using the PROMIS Alcohol Negative Consequences scale; and alcohol-related withdrawal is measured using the CIWA-AR scale. The PACS and PROMIS Alcohol Negative Consequences are used as efficacy endpoints, while the ACQ-SF-R and CIWA-AR scales are safety endpoints.

The ACQ-SF-R contains 12-items adapted from the 47-item ACQ-NOW developed by <u>Singleton et al (1994)</u> to assess craving for alcohol among alcohol users in the current context (right now). Items 3, 8, and 11 are reverse keyed. A general craving index is derived by summing all items and dividing by 12. If an item is missing, then the number of items is reduced by the number missing, and the sum is only the sum of the answered items. At least 10 items must be endorsed for the general craving index of ACQ-SF-R to be considered non-missing (i.e., scored).

The PACS is a five-item self-administered instrument for assessing craving (<u>Flannery-1999</u>). Frequency, intensity, and duration of thoughts about drinking are assessed along with ability to resist drinking. The final item asks the responder to provide an average rating of his/her craving over the course of the past week. The questions on the PACS use descriptors coupled with numerical ratings ranging from 0 to 6. The items are summed for a total score.

PROMIS Alcohol Negative Consequences scale is for negative consequences from alcohol use. The short form of the PROMIS Alcohol Negative Consequences questionnaire will be used to assess outcomes of alcohol use over the past 30 days (<u>Pilkonis-2013</u>).

#### The 7 PROMIS items include:

- Drinking created problems between me and others
- I disappointed others when I drank
- I was unreliable after I drank
- Others complained about my drinking
- I used poor judgment when I drank
- I said or did embarrassing things when I drank
- I had trouble getting things done after I drank

Each item is rated on a 5 point scale including: Never (1), Rarely (2), Sometimes (3), Often (4), and Almost Always (5) for the past 30 days. A subject's total score is converted to a T-score using scoring table provided by NIH PROMIS.

The CIWA-AR modified telephone version is an adaptation for telephone administration of the CIWA-AR a brief 10-item measure used to provide a quantitative index of the severity of the alcohol withdrawal syndrome (Sullivan et al-1989). The CIWA-AR has been used both in clinical and research applications and has demonstrated both reliability and validity (Sellers et al-1992, Stuppaeck et al-1994). The total score is the sum of the individual item scores. Since this is an interview scale, no missing items are anticipated. A score  $\geq$  10 is considered an indication that the subject is undergoing alcohol withdrawal.

#### **5.4. Mood**

Mood will be measured with the POMS.

The POMS measures dimensions of affect or mood (McNair and Heuchert-2005). It consists of 65 adjectives to which the subject responds according to a 5-point scale ranging from "not at all (0)" to "extremely (5)." Six subscale scores will be computed for items grouped as follows: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. A Total Mood Disturbance score will also be computed which consists of the sum of Tension-Anxiety, Depression-Dejection, Anger-Hostility, Fatigue-Inertia, and Confusion-Bewilderment scores then subtracting the Vigor-Activity subscale score. A missing value within a subscale will be replaced by the average score of the answered items within the subscale; if 2 or more items within a subscale are missing then the entire subscale is missing (Macefield et al-2010).

## 5.5. Sleep Quality

Sleep quality will be measured using the PSQI. The PSQI is a 19-item questionnaire (<u>Buysse et al-1989</u>). The addition of all the scores permits an analysis of the subject's overall sleep experience in the past 30 days. The lower the overall score, the better the person sleeps. A score  $\geq 5$  is indictive of a sleep disturbance. If any of the items is missing, then the entire form is missing for that evaluation (PSQI website).

#### 5.6. Cigarette Smoking Quantity-Frequency and Nicotine Use Questionnaire

A smoking quantity frequency and nicotine use interview will include 3 questions to assess nicotine use via cigarette smoking or via other products during the study: 1) Over the past week, on how many days did you smoke cigarettes?; 2) On the days you smoked during the past week, how many cigarettes did you smoke on average?; and 3) Over the past week, on how many days did you use other nicotine products (ex. chew, cigars, cigarellos, e-cigarettes, vape, gum, patch, etc...)? At baseline subjects that answer "0" to question #1 are considered non-smokers for the study. Cigarettes per week is the answer to question #1 multiplied by the answer to question #2. At baseline, subjects who report smoking (question #1) or the use of other nicotine product (question #3) will be considered nicotine users. The responses to questions #1 and #3 will be used to calculate the percentage of subjects abstinent from nicotine use among nicotine users. No imputation for missing values will be used.

#### 6. HYPOTHESES TO BE TESTED

#### 6.1. Primary Efficacy Endpoint

Subjects treated with ANS-6637 600 mg/day will report significantly lower VAS craving ratings in response to *in vivo* alcohol cues during human lab testing than ANS-6637 200 mg/day and placebo-treated subjects. Subjects treated with ANS-6637 200 mg/day will have significantly lower VAS craving ratings in response to *in vivo* alcohol cues than placebo-treated subjects.

The hypotheses for the confirmatory secondary endpoints for the cue reactivity sessions are the same as for the primary endpoint.

#### 6.2. Secondary Efficacy Endpoints

In the same dose-response manner, it is hypothesized that, during the last 4 weeks of the treatment period, the ANS-6637 groups, as compared to the placebo group, will:

- 1. Increase the percentage of subjects with no heavy drinking days. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
- 2. Increase the percentage of subjects abstinent from alcohol
- 3. Increase the percentage of subjects with at least a WHO 2-level decrease in alcohol consumption
- 4. Increase the percentage of subjects with at least a WHO 1-level decrease in alcohol consumption
- 5. Increase the percentage of days abstinent per week
- 6. Decrease the percentage of heavy drinking days per week
- 7. Decrease the percentage of very heavy drinking days per week
- 8. Decrease the weekly mean number of drinks per week
- 9. Decrease the weekly mean drinks per drinking day
- 10. Decrease the weekly mean cigarettes smoked per week among smokers
- 11. Increase the percentage of subjects abstinent from nicotine use among subjects who used any nicotine products in the week before randomization
- 12. Decrease the mean alcohol craving score (PACS)
- 13. Decrease the mean PSQI score
- 14. Decrease total mood disturbance (POMS)
- 15. Decrease in alcohol negative consequences (PROMIS)

#### 7. SAMPLE SIZE CONSIDERATIONS

Analysis of covariance with clinical site and baseline cue as the covariates will be used to model the primary outcome – the VAS craving score for the first alcohol cue. Statistical power was estimated using [PASS 13] with the following parameters. The treatment effect parameter—a maximal 3-point medication-placebo difference on the strength of VAS craving in response to the alcohol cue—was obtained from Roberts (2017), which used a similar cue reactivity paradigm. The mean values on this outcome at Week 2 are assumed to be 11 for 600 mg ANS-667, 12.5 for 200 mg ANS-667, and 14 for placebo and a standard deviation between subjects of 4. Clinical site and the baseline VAS craving for the alcohol cue were assumed to have correlations of 0.13 and 0.39, respectively, with the primary outcome. These correlations, coupled with assumed standard deviations for site and baseline VAS craving for the alcohol cue of 0.82 and 4, respectively, yield explained variation of 26%. These assumptions, with a sample size of 27 subjects per arm (81 total subjects), provides 82% statistical power with a 0.05 two-sided significance level. Using the Tukey test to adjust for the pairwise treatment arm comparisons reduces the power to 81% with a family-wise Type 1 error of 0.05 in 1000 simulations given the above assumptions.

#### 8. DATA QUALITY ASSURANCE

Data quality assurance will start with training of clinical investigative staff on data collection and assessment procedures including a Manual of Operations that describes what data to collect and procedures for completion of eCRFs. Completed eCRFs will be reviewed by Fast-Track Drugs and Biologics clinical monitors on a regular basis throughout the trial by comparison against the source documents.

Study data will come from the eCRFs, TLFB spreadsheets, coded AEs, AiCure Drug Compliance system outputs, genetics testing lab spreadsheets and PK drug levels from the PK lab spreadsheetseCRFs for this study were created using an electronic data management system (EDMS) based on IBM clinical development system. eCRFs were created using an established data dictionary for each variable including the field name, field type, field attributes, and coding for variables. Range checks, alpha-numeric requirements, and null/not null parameters were programmed as applicable. The back end database application is Oracle. Data entered into the EDMS system will be reviewed by Fast-Track clinical monitors and data managers. If incomplete or inaccurate data are found, the data will be queried in the system for site staff to address. The site will resolve data inconsistencies and errors using the EDMS with full audit trail of corrections being maintained within the system. Corrections and changes to the data will be reviewed by Fast-Track clinical monitors and data managers. TLFB spreadsheets have a double data entry check system and additionally, Fast-Track staff will verify the data entries with the drinking calandar to verify the correct percentages of alcohol by volume. QA review of laboratory data outputs is the responsibility of the individual testing laboratories; however, Fast-Track staff will verify that there is a result reported for each specimen that was recorded in the database as being collected. Coded AEs will be cross checked by a second trained MedDRA coder

Additional edit checks will be written to detect anomalies in the database. These checks will address inconsistencies (within visits, across visits), invalid/unusual values, missing values, and protocol violations. Edit checking will be validated on test data or actual clinical trial data. In addition to programmed edit checks, quality control examination of data will also be performed on reviews of data listings.

#### 9. STATISTICAL CONSIDERATIONS

#### 9.1. General Considerations

For descriptive purposes, dichotomous and categorical variables will be presented as number of observations and percentages; continuous variables will be given as means, standard deviations (SD), median, miniumum (min) and maximum(max). Statistical tests will be two-tailed at a 0.05 Type I error rate. P-values for the primary and secondary endpoints of < 0.05 will be considered statistically significant. Endpoint data will also be screened for outliers and skewness. Appropriate non-parametric tests will be used to compare treatment groups on continuous baseline characteristics that are not normally distributed. Continuous endpoint data that are not normally distributed will be transformed using either a square root, logarithmic, or inverse transformation, the selection of which is determined by skewness and kurtosis statistics with values closest to zero. Cohen's d will be used to calculate the effect size for means and Cohen's h or odds ratios will be used to calculate the effect size for proportions. Descriptive statistics — mean, SD, median, min and max — of all endpoint data will be provided for each assement point or summarized at each week for drinking endpoints. All data will be presented in listings.

# 9.2. Participant Accountability and Protocol Deviations

A summary will be prepared to show dropouts/retention over time in each group, along with the reason for early discontinuation. The number of missing observations will be presented between groups. Protocol deviations will be presented as summaries by type of deviation.

## 9.3. Demographics and Other Baseline Characteristics

Summaries of the characteristics of the subjects in each of the study groups at baseline will be prepared for the mITT, and evaluable analysis sets. Demographic characteristics (e.g., age, gender, race, ethnicity, marital status, employment, and education) and other baseline characteristics including ALDH2 genetics testing results, screening cue session VAS scale scores and ACQ-SF-R pre and post session score, mood scales (e.g., POMS total and subscale scores), PSQI, and drinking goal, MINI AUD scores and other DSM-5 diagnoses will be summarized by treatment group for the mITT and evaluable subjects. ANOVA or chi-square tests will be used on baseline characteristics to test the hypothesis of effective randomization. Imbalance in any of these factors is an indication of ineffective randomization which may bias the results observed on any of the endpoints.

Baseline drinking parameters in the 28-days prior to the start of screening, age started drinking regularly, medical treatments for drinking in the past year, and other services used for alcohol problems in the past 4 weeks prior to consent will be summarized by treatment group for the mITT subjects. ANOVA will be used for baseline drinking parameters to test the hypothesis of effective randomization. The number and percentage of subjects with mild, moderate and severe symptoms of AUD and summary statistics for total number of symptoms will also be presented.

The quantity of cigarettes smoked per week in the week prior to randomization will be presented for those subjects who reported any smoking. The numbers and percentages of subjects who report other nicotine product use at baseline, any nicotine use, and who test positive for THC will also be presented. Because smoking, any nicotine use, and positive THC are subsets and are not

controlled by randomization, balance across treatment groups will be assessed using ANOVA and chi-square tests.

Baseline drinking-associated consequences (CIWA-AR and PROMIS Alcohol Negative Consequences scores) and drinking-associated-craving (PACS) total score and subscales will be summarized in the tables. ANOVA will be used to test for balance across the treatment groups and evaluate the hypothesis of ineffective randomization.

Continuous variables will be summarized using means, standard deviations, medians, minimum, and maximum values. Categorical variables will be summarized using counts and percentages.

## 9.4. Efficacy Analysis

#### 9.4.1. Primary Analysis of the Primary Efficacy Endpoint

Each subject will have an initial alcohol cue for "strength" of craving score from the VAS that is the primary endpoint. Analysis of covariance (ANCOVA) with the "strength" of alcohol craving value as the dependent variable and the pretreatment "strength" of alcohol craving score from the first alcohol cue as an independent fixed effect. Clinical site will also be included as an independent factor. There are 3 comparisons (ANS-6637 600 mg vs placebo; ANS-6637 200 mg vs. placebo; ANS-6637 600 mg vs. ANS-6637 200 mg) and Tukey's method will be used to maintain a family-wise 0.05 significance level.

No imputation for missing endpoint data will be performed.

### 9.4.2. Confirmatory Secondary Endpoints

There are 3 additional VAS craving questions and a beverage liking question asked during the human lab session. Each of these questions will be analyzed in the same manner as listed in Section 9.4.1. Tukey's method will be used within question and not across questions. An overall mean of the 4 VAS craving items will also be analyzed similarly for just the alcohol beverage cue. The difference between the first alcohol cue and water cue for each VAS item will be computed at both the pre and post treatment time points. The difference values for each VAS item and the average difference will be analyzed similarly to the primary endpoint.

#### 9.4.3. Analysis of the Secondary Efficacy Endpoints

Secondary efficacy endpoints will also be analyzed based on data collected during the last 4 weeks of the maintenance period (Weeks 2 through 5), including TLFB and other questionnaire data assessed at Week 6 that reflect data collected during this period.

In general, every continuous secondary efficacy endpoint is analyzed using a repeated measures mixed effects model where subjects are random effects; factors and covariates are fixed effects. The analyses will be performed using SAS PROC MIXED procedure. The information criterion is requested from every mixed effects model. Subjects are treated as a class variable and not continuous. The week (Weeks 2 through 5), treatment group, and clinical site are also treated as class variables

The primary analysis model for all continuous endpoints is:

• Appropriately transformed endpoint = treatment + week + treatment\*week + clinical site + baseline equivalent of endpoint + other covariates (identified in Section 9.4.4)

This model will also be created for the untransformed endpoint. The solution statement from SAS PROC MIXED is requested to provide the solution for the fixed effects parameters. A REPEATED statement specifies that values are repeated each week and subjects are nested within treatment group. The covariance structure is specified.

The selection of the covariance structure is performed using a simple repeated mixed effects model that includes treatment group as the only fixed effect and subject nested within treatment group as the only random effect. The covariance structure for each continuous secondary endpoint is selected from autoregressive, compound symmetry, Toeplitz, and unstructured. The Akaike Information Criterion (AICc) corrected for a finite sample is obtained from each of the four models for the four possible covariance structures to determine model fit. The smallest (minimum) AICc associated with one of the covariance structure is selected and the difference for each of the other three covariance structures are calculated. A graph is produced of the model fit statistics and relative difference for the four possible covariance structures. The graphs across the continuous endpoints are compared to determine which covariance structure will be selected for all continuous endpoints or if one or more models need different covariance structures.

Results based on the primary analysis model and the model of the untransformed endpoint will be presented in tabular form. The overall least squares means and least square means for each time point along with the 95% confidence intervals (CI) will be presented for the untransformed endpoint only, while two-tailed p-values and Cohen's d will be presented for both the untransformed and transformed data. Inference and Cohen's d will be based upon the results using appropriately transformed data. Graphs of all secondary endpoints will be produced.

## 9.4.3.1. Secondary Drinking Endpoints

Percentage of days abstinent per week, percentage of subjects abstinent, percentage of heavy drinking days per week, percentage of very heavy drinking days, weekly mean number of drinks per week, and weekly mean number of drinks per drinking day will be analyzed using the mixed effects model specified in Section 9.4.3. Covariates for these models will be identified as in Section 9.4.4.

Percentage of subjects with a WHO 1-level decrease, and WHO 2-level decrease in alcohol consumption risk category will be analyzed during the last 4 weeks of the maintenance period (Weeks 2 through 5) using a logistic regression model. Covariates for the logistic regression will be identified as in Section 9.4.4. 2x2 contingency tables will report the WHO 1-level decrease, and WHO 2-level decrease along with Cohen's h, odds ratios and 95% CIs. The Wald statistic will be used to test for treatment differences.

No adjustment for multiple comparisons and no imputation will be used for these endpoints.

#### 9.4.3.2. Alcohol Consequences and Craving Scales

The PACS is assessed weekly and will be analyzed similarly to the drinking endpoint (Section 9.4.3.1). PROMIS alcohol negative consequences scale is assessed at baseline and Study Week 6

which will be used for the secondary endpoint. Analysis of covariance will be used to analyze the PROMIS scale similarly to the primary endpoint (Section 9.4.1).

No imputation or multiplicity adjustment will be used for this endpoint.

# 9.4.3.3. Smoking and Any Nicotine Use

The mean number of cigarettes smoked in the past week is measured at weekly. The sample is the mITT subjects who smoked at baseline. The data will be analyzed as described in Section 9.4.3. Covariates for this endpoint will be identified in Section 9.4.4. Amount of other nicotine products is not captured, only number of days of use of other nicotine products. The analysis of days of use in subjects using other nicotine products at baseline will use the same method as cigarettes smoked. In addition, 2 tables will examine the number of subjects that are abstinent from cigarettes and any nicotine product use. There will be one logistic regression, if there are sufficient number of subjects abstaining from nicotine use, with abstaining as the dependent variable and covariates as described in Section 9.4.4. No imputation will be used for these endpoints.

## 9.4.3.4. Sleep and Mood Scales

The PSQI total score POMS 6 subscales and total disturbance score are continuous variables. The secondary endpoints for the POMS is assessed at Study Weeks 4 and 6. The PSQI total score is assessed at Week 6. The data will be analyzed as described in Section 9.4.3. Covariates for these models will be identified as in Section 9.4.4.

No imputation or multiplicity adjustment will be used for these endpoints.

#### 9.4.4. Covariate Adjustment for the Analysis of Secondary Efficacy Endpoints

Covariates for continuous secondary efficacy endpoints include the baseline equivalent of the endpoint, clinical site, treatment, time and the treatment by time interaction. Additional covariates for the secondary efficacy endpoints may include baseline characteristics with a theoretical and/or empirical basis for a relationship with a particular secondary endpoint. Such characteristics may include, but are not limited to, drinking goal (stop drinking versus reduce drinking but not stop), age, and baseline alcohol craving scale total score. Prior to the unblinding of the data, matrices of correlations between these baseline characteristics and each of the secondary efficacy endpoints, pooled across blinded treatment assignment, will be produced (using Pearson for continuous variables, Spearman for categorical outcomes). Selection of baseline variables to include as covariates in the models will be based on consideration of the following criteria: at least modest correlation with outcome (i.e.,  $r \ge 0.20$ ) and clinical expertise. Each endpoint may have a unique set of covariates. Care is taken to only select a limited number of covariates such that the models are not over fitted.

Covariates for the dichotomous secondary endpoints, percentage of subjects abstinent, WHO 1-level risk category decrease, and WHO 2-level risk category decrease in alcohol consumption, will use phi correlation with dichotomous variables, chi-square statistic for categorical variables, and biserial correlation. Fewer covariates for the logistic regression may be used depending upon the number of events. If the number of events permits the inclusion of a baseline drinking covariate, the percentage of days abstinent will be used as the covariate for the percent subjects abstinent endpoint and the percent heavy drinking days will be used as the covariate for the Statistical Analysis Plan: Protocol HLAB-002, Version 1.0 Dated: 16Mar2020

percent subjects with no heavy drinking days endpoint; however, no baseline drinking covariate will be employed for the endpoint, percent subjects with a WHO decrease in alcohol consumption, as this endpoint already adjusts for baseline drinking in its calculation.

## 9.5. Handling of Missing Data

The primary endpoint of craving cannot be imputed; likewise, for the other craving questions given during the human lab session. Secondary endpoints analyzed with mixed effects or logistic regression models are capable of handling missing data, so no imputation will be utilized. PROMIS scores are analyzed using ANCOVA which cannot handle missing data; therefore, only subjects with an assessment during the treatment period will be used and no imputation.

#### 9.6. Safety Analysis

#### 9.6.1. Adverse Events

There are both voluntary and elicited AEs. Voluntary AEs will be coded using the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be grouped by system, organ, and class (SOC) and preferred term (PT) designation. The severity, frequency, and relationship of AEs to investigational product will be presented by SOC and PT groupings. Subjects asked questions about appetite, heat sensation, and increased heart rate will be reported separately. All subjects that answer "yes" to any of the elicited questions will have a separate listing presenting their adverse events. AEs will be presented by ALDH2 deficient and ALDH2 non-deficient patients and by subjects who did or did not take any drugs with potential for drugdrug interactions including proton pump inhibitors, histamine-2 antagonists,. OATP1B1 and OATP1B3 transporters, OAT1 and OAT3 transporters, MATE1, MATE-2K, and OCT2 transporters, P-gp transporter thhibitors, and BCRP transporters. Listings of each individual AE including start date, stop date, severity, relationship, outcome, and duration will be provided. Each AE (based on PT) will be counted once only for a given study subject. If the same AE occurred on multiple occasions, the highest severity will be assumed. Thus, study subjects are not counted multiple times in a given numerator in the calculation of frequencies for a specific AE. C-SSRS reports of suicidality or suicidal ideation will be reported as AEs and analyzed as AEs if the investigator determines after an interview with the subject, that the responses are consistent with suicidal ideation or attempt.

## 9.6.2. Clinical Laboratory and Point of Care Tests

For clinical laboratory data, descriptive statistics will be generated for all tests performed at screening and at each clinic visit. If a laboratory analysis is repeated, the last measurement performed prior to the clinic visit will be used in the summary statistics for that clinic visit. If an unscheduled clinical laboratory visit occurs prior to a scheduled visit that is missed due to dropout, then the unscheduled visit will be used in the summary statistics for the missed scheduled clinical visit. If an unscheduled clinical laboratory visit occurs between two scheduled clinical visits, then the data from the unscheduled visit only be presented in the listings and not in summary statistics. In addition, at each post-randomization clinic visit descriptive statistics for change from baseline will be generated. Laboratory values will be plotted as mean ± standard error over time. All laboratory measurements will be presented in the listings.

Number and percentage of positive urine drug tests and pregnancy tests for screening visits and all treatment and follow-up visits will be tabulated. Results of all urine drug tests and pregnancy tests will be presented in the listings. The percentage of subjects with a positive urine drug test at any time post start of treatment will also be presented by test type and treatment group.

# 9.6.3. Vital Signs, ECG, and Body Weight

Vital signs will be presented as summary statistics and change from baseline. The percentage of ECG results considered abnormal and clinically significant will be provided. Body weight will be presented as summary statistics and change from screening. Vital signs, ECG results, and weight measurements for all visits will be presented in the listings.

#### 9.6.4. CIWA-AR Scores

The number and percentage of subjects who reported CIWA-AR scores  $\geq 10$  at any time after the start of dosing will be presented.

#### 9.6.5. ACQ-SF-R Scores

Summary statistics for ACQ-SF-R raw scores prior to after each cue session will be presented. The number and percentage of subjects with a higher ACQ-SF-R score post each cue session will be provided by treatment group.

## 9.7. Drug Exposure and Retention Analyses

Drug exposure will be presented for each treatment group as the mean number of tablets taken by week and overall through AiCure during the entire treatment phase. The analysis will include the total number of tablets taken and the percent compliance. AiCure data will also be used for the number subjects receiving reminder intervention (phone calls, texts, or in person visits). In addition, medication bottles are returned and the number of tablets remaining in those bottles are documented. It is assumed that the missing tablets would have been consumed. Compliance will also be evaluated by determining the proportion of subjects who were prescribed ANS-6637, reported taking ANS-6637 (by AiCure assessment), and had a plasma sample with detectable GS-548351, the active moiety of ANS-6637. Compliance by GS-548351 plasma levels will be reported as number and percentage of subjects with a level above the limit of detection at each time point. Descriptive statistics of plasma levels will also be provided.

#### 9.8. Blood Alcohol Content

The number and percent of subjects at any clinic visit that have a BAC > 0 will be tabulated. All BAC measurements will be presented in the listings.

# 9.9. Exploratory Analyses

#### 9.9.1. Value of the Second Alcohol Cue

Each subject will be presented with a water cue followed by an alcohol cue then followed by a second alcohol cue. Each VAS question will be asked after each cue. To determine whether there is any difference with the 2<sup>nd</sup> alcohol cue at baseline the combined data across treatment groups will be used. Paired t-tests will be used for each question to test the hypothesis that no difference

in response between the first and second alcohol cue. This analysis will be performed at Week 2 lab session.

If there is a difference between the first and second alcohol cue then the primary endpoint analysis as indicated in Sections 9.4.1 and 9.4.2 will be repeated with the 2<sup>nd</sup> alcohol cue VAS in addition to the 1<sup>st</sup> alcohol cue. Only those VAS questions that showed a difference between the first and second alcohol cue will be examined.

#### 9.9.2 Supplemental Exploratory Analyses

Two additional exploratory analyses are defined as: 1. Explore moderators of the treatment effect on primary and secondary outcomes; 2. Examine the relationship between cue-reactivity craving in the lab and naturalistic secondary outcomes. These two exploratory endpoints will not be analyzed at the same time as the primary and secondary endpoints.
#### 10. VALIDATION OF PROGRAMMING CODE

All SAS codes used to generate tables and listings will be validated and reviewed before being finalized. The validation process will be used to determine that the numbers are produced by a statistically valid method and that the execution of the computations is correct. Qualified personnel who have not previously been involved in the production of the original programming codes will perform the validation procedures. Methods of validation include independent programming and comparison to data listings. Tables will be reviewed for accuracy, consistency with this plan, consistency within tables, and consistency with corresponding output. Once validation is complete, a quality control reviewer will perform a final review of the documents for accuracy and consistency. Upon completion of validation and quality review procedures, all documentation will be collected and filed in the study documentation files at Fast-Track.

#### 11. REFERENCES

Aubin HJ, Reimer J, Nutt DJ, Bladstrom A, Torup L, Francois C, Chick J. Clinical relevance of as-needed treatment with nalmefene in alcohol dependent patients. Eur Addict Res. 2015;21:160–68.

Buysse, D. J., Reynolds, C. F., 3rd, Monk, T. H., et al. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989;28:193-213.

Carey KB. Reliability and validity of the time-line follow-back interview among psychiatric outpatients: a preliminary report. Psych Addic Behav. 1997;11, 26-33.

Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res 1999;23:1289-95.

Macefield RC, Metcalfe C, Lane JA, Donovan JL, Avery KNL, Blazeby JM, Down L, Neal DE, Hamdy FC, Vedhara K. Impact of prostate cance testing: evaluation of the emotional consequences of a negative biopsy result. Br J Cancer 2010;102:1335-1340.

Mason BJ, Light JM, Williams LD, Drobes DJ. Proof-of-concept human laboratory study for protracted abstinence in alcohol dependence: Effects of gabapentin. Addict Biol. 2009;14:73-83.

Mason BJ, Quello S, Goodell V, Shadan F. Gabapentin treatment for alcohol dependence. JAMA. 2014;174:70-77.

McNair DM, Heuchert JWP. Profile of Mood States (POMS) Multi-Health Systems, Tonawanda, NY. 2005.

Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. 1996;49:1373-1379.

Pilkonis PA, Yu L, Colditz J, Dodds N, Johnston KL, Maihoefer C, Stover AM, Daley DC, McCarty D. Item banks for alcohol use from the Patient-Reported Outcomes Measurement Information System (PROMIS): use, consequences, and expectancies. Drug Alcohol Depend. 2013;130:167-77.

Roberts W, Harrison ELR, McKee S. Effects of varenicline on alcohol cue reactivity in heavy drinkers. Psychopharmacology (Berl). 2017;234:2737-2745.

Sellers EM, Sullivan JT, Somer G, Sykora K. Characterization of DSM-III-R criteria for uncomplicated alcohol withdrawal: proposal for a diagnostic inventory and revised withdrawal scale. In Naranjo, C. A. and Sellers, E. M. (Eds.) Novel pharmacological interventions for alcoholism. New York (pp. 369-71). 1992.

Singleton EG, Tiffany, ST, Henningfield JE. Development and validation of a new questionnaire to assess craving for alcohol. In: Harris LS (ed) *Problems of Drug Dependence, 1994; Proceedings of the 56<sup>th</sup> Annual Scientific Meeting, The College on Problems of Drug Dependence, Inc.* National Institute of Drug Abuse Research Monograph Series. Vol. 153. Rockville, MD 1995. p. 289.

Sobell LC, Sobell MB, Leo GI, Cancilla A. Reliability of a timeline method: assessing normal drinkers' reports of recent drinking and a comparative evaluation across several populations. Br J Addict. 1988;83:393-402.

Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend 1996;42:49-54.

Stuppaeck CH, Barnas C, Falk M, Guenther V, Hummer M, Oberbauer H, Pycha R, Whitworth AB, Fleischhacker WW. Assessment of the alcohol withdrawal syndrome--validity and reliability of the translated and modified Clinical Institute Withdrawal Assessment for Alcohol scale (CIWA-A). Addiction. 1994;89:1287-92.

Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-AR). Br J Addict. 1989;84:1353-7.

World Health Organization (WHO): International Guide for Monitoring Alcohol Consumption and Related Harm. Geneva, WHO, 2000. Available at: http://whqlibdoc.who.int/hq/2000/who\_msd\_msb\_00.4.pdf.

- 12. TABLE, LISTING, AND FIGURE SHELLS
- **12.1.** Tables
- 12.1.1. Subject Disposition, Participation, Compliance

 Table 1:
 Subject Disposition - All Randomized Subjects

| | | Т | reatment Group | | |
|---|---|---|---|---|---|
| | Placebo | ANS-6637-<br>200mg | ANS-6637-<br>600mg | Total | |
| | n (%) | n (%) | n (%) | n (%) | p-value <sup>1</sup> |
| Number of Subjects Consented | | | | XX | |
| Number of Subjects Screen Failed | | | | XX | |
| Number of Subjects Randomized | XX | XX | XX | XX | 0.xxx |
| Number of Subjects Randomized not Receiving Study Drug | x (xx.x) | x (xx.x) | x (xx.x) | x (xx.x) | 0.xxx |
| Number of mITT Subjects | xx (xx.x) | xx (xx.x) | xx (xx.x) | xxx (xx.x) | 0.xxx |
| Number of Completed <sup>2</sup> Subjects | xx (xx.x) | xx (xx.x) | xx (xx.x) | xxx (xx.x) | 0.xxx |
| Number of Evaluable Subjects | xx (xx.x) | xx (xx.x) | xx (xx.x) | xxx (xx.x) | 0.xxx |
| Number of Subjects Discontinuing Medication, Remaining in Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Number of Subjects Discontinuing Medication, Drop out of Study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx |
| Reason for Early | | | | | |
| Lost to follow up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Died | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Logistical or practical reasons | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Lack of perceived efficacy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Absent from the protocol due to confinement in a controlled environment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Determined after randomization to be ineligible | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

| Subject withdrew consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|--------------------------|-----------|-----------|-----------|-----------|
| Clinical deterioration | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Prefer another treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol noncompliance | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other reason | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Notes: ¹ p-value from chi-square test (c), and Fisher's exact test (f). Fisher's exact test is used when any expected number in a cell for a specific row is less than 5.

<sup>2</sup>Completed is defined as completing the full intervention phase (Weeks 2-5) of the study making the subject available for all endpoint analyses

Programmer Notes: The discontinuation reasons are as given on the CRF. Include only the reasons actually used for the subjects in the study. If a subject discontinued, but the specific reason is missing, include 'Missing' as a row in the table. Use the order of discontinuation reasons as presented on the CRF page.

**Table 2:** Exposure to Investigational Products Using AICure Data – mITT Subjects

| | | Pla | acebo | | | AN | S-6637 | 200mg | | ANS-6637 60 | ANS-6637 600mg | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean<br>(SD³) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) | p-value <sup>1</sup> |
| Week 1 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 2 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 3 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 4 | XX | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Week 5 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |
| Total Dose <sup>2</sup> | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | 0.xxx |

<sup>&</sup>lt;sup>1</sup> p-value from F-test from ANOVA

**Table 3:** Total Exposure to Investigational Products Using AICure Data – Evaluable Subjects

Same as Table 2 only using evaluable subjects

<sup>&</sup>lt;sup>2</sup> Dose is the total number of capsules taken

<sup>&</sup>lt;sup>3</sup> SD is standard deviation

## Table 4: Compliance to Investigational Products Using AICure Data – mITT Subjects

Same analysis as Table 2 using compliance rather than dose. Compliance is the number of capsules taken/number of capsules prescribed.

### Table 5: Compliance to Investigational Products Using AICure Data – Evaluable Subjects

Same analysis as Table 4 using evaluable subjects

**Table 6:** AiCure Interventions mITT Subjects

| | | Placebo | ANS 6 | 637 200 mg | ANS 6637 600 mg | |
|---|---|---|---|---|---|---|
| | N | # Receiving ≥ 1 | N | # Receiving ≥ 1 | N | # Receiving ≥ 1 |
| Interventions <sup>1</sup> | XX | XX | XX | xx | xx | XX |

<sup>&</sup>lt;sup>1</sup> Interventions includes texts, emails, and phone calls

## Table 7: AiCure Interventions – Evaluable Subjects

Same as Table 6 only using evaluable subjects

**Table 8:** Summary of GS-54851 Blood Levels – ANS6637 Groups (mITT Subjects)

| | | ANS | 5-6637 200mg | | | ANS-6637 600mg | | |
|---|---|---|---|---|---|---|---|---|
| | N | % > LLD <sup>1</sup> | Mean (SD <sup>2</sup> ) | (Min-Max) | N | % > LLD | Mean (SD) | (Min-Max) |
| Week 2 | xx | XX.X | xx.x (xx.x) | (xx.x-xx.x) | XX | XX.X | xx.x (xx.x) | (xx.x-xx.x) |
| Week 4 | xx | XX.X | xx.x (xx.x) | (xx.x-xx.x) | xx | XX.X | xx.x (xx.x) | (xx.x-xx.x) |

<sup>&</sup>lt;sup>1</sup> LLD is lowest level of detection

## Table 9: Summary of GS-54851 Blood Levels – ANS6637 Groups (Evaluable Subjects)

Same as Table 8 only using evaluable subjects.

<sup>&</sup>lt;sup>2</sup> SD is standard deviation

Table 10: AiCure Report of ANS-6637 Versus GS-5851 Blood Levels – mITT Subjects

| | | Pill Count Ir<br>Taken | idicates Drug | | |
|---|---|---|---|---|---|
| Timing | Blood level<br>Indicates Drug<br>Taken <sup>a</sup> | Yes, n (%) | No, n (%) | p-value <sup>b</sup> | kappa <sup>c</sup> |
| Week 2 | Yes | | | | |
| | No | | | | |
| Week 4 | Yes | | | | |
| | No | | | | |
| Overall | Yes | | | | |
| | No | | | | |

<sup>&</sup>lt;sup>a</sup> Blood level of ≥80 ng/mL indicates drug taken

note this will be repeated for ANS-6637 600 mg

b Chi-square test for independence

c Kappa test for agreement

Table 11: AiCure Report of ANS-6637 Versus GS-5851 Blood Levels – Evaluable Subjects

Repeat of Table 10 using evaluable subjects

**Table 12:** Exit Interview – mITT Subjects

| | Placebo | ANS-6637<br>200 mg | ANS-6637<br>600 mg | Total | |
|---|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Did you think you were receiving the study drug or the placebo? | | | | | 0.xxx |
| Placebo | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Study Drug | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Don't know; No idea | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| What is your desire to please people? | | | | | 0.xxx |
| More than average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | Placebo | ANS-6637<br>200 mg | ANS-6637<br>600 mg | Total | |
|---|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Less than average | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Take the study drug again, for more than 5 weeks? | | | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Did you limit your drinking<br>because of flushing (a heat<br>reaction or facial redness)? | | | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Did you limit your drinking beca | use of nausea or of | ther effects? | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | Placebo | ANS-6637<br>200 mg | ANS-6637<br>600 mg | Total | |
|---|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Did your friends or family notice flushing? | | | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| If your friends or family noticed flushing, did this change your drinking? | | | | | , |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Did you ever miss a dose of medication to avoid these effects? | | | | | <u> </u> |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | Placebo | ANS-6637<br>200 mg | ANS-6637<br>600 mg | Total | |
|---|---|---|---|---|---|
| Question | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Did you use any other services during the study to help you reduce drinking? | | | | | 0.xxx |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Refuse to answer | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

¹ p-value from chi-squared test (c) unless one of the cells expected is less than 5 then Fisher's exact test is used (f). Refuse to answer is not included in statistical test.

**Table 13:** Exit Interview – Evaluable Subjects

Same as Table 12

**Table 14:** Dropouts by Treatment Group and Week – mITT Subjects

| | Placebo | | ANS-6637 200<br>mg | | ANS | ANS-6637 600 mg | | Total | |
|---|---|---|---|---|---|---|---|---|---|
| Study<br>Week <sup>2</sup> | n | Cumulative<br>n (%) | n | Cumulative<br>n (%) | n | Cumulative<br>n (%) | n | Cumulative<br>n (%) | p-value <sup>1</sup> |
| Week 1 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 2 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 3 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 4 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 5 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |
| Week 6 | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | 0.xxx |

 $<sup>^{1}</sup>$  Fisher's exact test is used since the frequencies are expected to be low

<sup>&</sup>lt;sup>2</sup>Subjects are considered dropouts when they stop providing TLFB and other data. Subjects that discontinue study drug but provide data are not considered dropouts.

Table 15: Number and Percent of Subjects Using Summary Drinking Questions after Discontinuing TLFB – mITT Subjects

| | Placebo | ANS-6637 200<br>mg | ANS-6637<br>200 mg | Total | |
|---|---|---|---|---|---|
| Study Week | n (%) | n (%) | n (%) | n (%) | p-value <sup>1</sup> |
| Week 3 | xx (xx.x) | XX | xx | xx.x% | 0.xxx |
| Week 4 | XX | xx | XX | xx.x% | 0.xxx |
| Week 5 | XX | xx | XX | xx.x% | 0.xxx |
| Week 6 | xx | xx | XX | xx.x% | 0.xxx |
| Overall | XX | XX | XX | xx.x% | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Fisher's exact test is used because frequencies are expected to be low

Note only rows with values above 0 will be presented

| 12.1.2. | Demographic and Baseline Characteristics |
|---------|------------------------------------------|

 Table 16: Demographic Characteristics - mITT Subjects

| | | ANS-6637 | ANS-6637 | | |
|---|---|---|---|---|---|
| Characteristic | Placebo | 200 mg | 600 mg | Total | p-value <sup>1</sup> |
| Age (years) | | | | | 0.xxx |
| N | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD <sup>2</sup> | XXX.XX | XXX.XX | XXX.XX | xxx.xx | |
| Median | XX | XX | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Gender | | | | | 0.xxx |
| N | | | | | |
| Male | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Female | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Race | | | | | 0.xxx |
| N | XX | XX | XX | XX | |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| African-American or Black | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Asian | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | | ANS-6637 | ANS-6637 | | |
|---|---|---|---|---|---|
| Characteristic | Placebo | 200 mg | 600 mg | Total | p-value <sup>1</sup> |
| American Indian or Alaskan Native | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ethnicity | | | | | 0.xxx |
| N | xx | XX | XX | XX | |
| Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not Hispanic or Latino | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Education (years) | | | | | 0.xxx |
| N | xx | XX | XX | XX | |
| Mean | xx.x | XX.X | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | |
| Median | xx | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx | xx) | (xx | |
| Marital Status | | | | | 0.xxx |
| Legally Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Living with Partner / Cohabitating | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Widowed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Separated | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | | ANS-6637 | ANS-6637 | | |
|---|---|---|---|---|---|
| Characteristic | Placebo | 200 mg | 600 mg | Total | p-value <sup>1</sup> |
| Divorced | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Never Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Employment | | | | | 0.xxx |
| Full-time > 35 hrs /week | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Part-time regular | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Part-time irregular | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Student | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Military Service | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unemployed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Retired/Disabled | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Homemaker | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| In controlled environment | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Annual Income | | | | | 0.xxx |
| \$0-\$15,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$15,001-\$30,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$30,001-\$45,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$45,001-\$60,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | | ANS-6637 | ANS-6637 | | |
|---|---|---|---|---|---|
| Characteristic | Placebo | 200 mg | 600 mg | Total | p-value <sup>1</sup> |
| \$60,001-\$75,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$75,001-\$90,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$90,001-\$105,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| \$105,001-\$120,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Greater than \$120,000 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| None given | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Occupation | | | | | 0.xxx |
| Executive of large business or major | | | | | |
| professional | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Manager of medium business or minor | | | | | |
| professional | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Administrator of large business, owner of small | | | | | |
| business, or semi-professional | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clerical or sales worker, technician | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Skilled worker | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Semi-skilled worker | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unskilled worker | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Unemployed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

| | | ANS-6637 | ANS-6637 | | |
|---|---|---|---|---|---|
| Characteristic | Placebo | 200 mg | 600 mg | Total | p-value <sup>1</sup> |
| Never worked | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not given | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

<sup>&</sup>lt;sup>1</sup>c = chi-squared test, f=Fisher's exact test, w=Wilcoxon signed rank test

 Table 17:
 Dichotomized Demographic Characteristics – mITT Subjects

| | | ANS-6637 | ANS-6637 | | |
|---|---|---|---|---|---|
| Characteristic | Placebo | 200 mg | 600 mg | Total | p-value <sup>1</sup> |
| Race/Ethnicity | | | | | 0.xxx |
| White | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| African-American or Black | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Hispanic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Education | | | | | 0.xxx |
| Less than High School | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| High School or Greater | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

<sup>&</sup>lt;sup>2</sup> SD is standard deviation

| | | ANS-6637 | ANS-6637 | | |
|---|---|---|---|---|---|
| Characteristic | Placebo | 200 mg | 600 mg | Total | p-value <sup>1</sup> |
| Marital Status | | | | | 0.xxx |
| Legally Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not Married | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Employment | | | | | 0.xxx |
| Unemployed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Employed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

<sup>&</sup>lt;sup>1</sup>c = chi-squared test, f=Fisher's exact test, w=Wilcoxon signed rank test

**Table 18:** Demographic Characteristics – Evaluable Subjects

Same as Table 16

Table 19; Dichotomized Demographic Characteristics – Evaluable Subjects

Same as Table 17

 Table 20:
 Screening Cue Reactivity – mITT Subjects

| | | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | N=xx | |
| Cue | Question | Statistic | | | | | |
| Water | Craving<br>Strength | | | | | | 0.xxx |
| | | Mean (SD <sup>2</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drinking makes things perfect | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drink now | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |

| | | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | N=xx | |
| | Turn down drink | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Average | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Alcohol 1 | Craving<br>Strength | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drinking makes<br>things perfect | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |

| | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | | N=xx | N=xx | N=xx | N=xx | |
| | Median | xx | XX | XX | xx | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drink now | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | xx | XX | xx | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Turn down drink | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | xx | XX | xx | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Average | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | xx | XX | xx | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |

| | | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | N=xx | |
| Alcohol 2 | Craving<br>Strength | | | | | | 0.xxxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Driking makes<br>things perfect | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drink now | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | xx | XX | xx | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Turn down drink | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |

| | | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | N=xx | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Average | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Alcohol1 -<br>Water | Craving<br>Strength | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drinking makes things perfect | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |

| | | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | N=xx | |
| | Drink now | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Turn down drink | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Average | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | XX | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Alcohol2 -<br>Water | Craving<br>Strength | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |

| | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | | N=xx | N=xx | N=xx | N=xx | |
| | Median | XX | XX | XX | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinking makes things perfect | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX | xx | XX | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drink now | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | xx | xx | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Turn down<br>drink | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | xx | xx | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |

| | | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|---|
| | | | N=xx | N=xx | N=xx | N=xx | |
| | Average | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Alcohol1 –<br>Alcohol2 | Craving<br>Strength | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drinking makes things perfect | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | | Median | XX | XX | XX | xx | |
| | | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| | Drink now | | | | | | 0.xxx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |

| | | Placebo | ANS-6637 200<br>mg | ANS-6637 600<br>mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| | | N=xx | N=xx | N=xx | N=xx | |
| | Median | xx | XX | XX | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Turn down<br>drink | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | XX | XX | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Average | | | | | | 0.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | xx | XX | xx | XX | |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |

<sup>&</sup>lt;sup>1</sup> ANOVA and F-test is used to examine balance across treatment groups

<sup>&</sup>lt;sup>2</sup> SD is standard deviation

# Table 21: Screening Cue Reactivity – Evaluable Subjects

Same as Table 20

 Table 22:
 Psychiatric Baseline Characteristics – mITT Subjects

| | Placebo | ANS-6637 300 mg | ANS-6637 600 mg | Total |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| DSM-5 Disorders | | | | |
| Depression | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suicidality | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Manic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hypomanic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bipolar | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Panic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Agoraphobia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Social Phobia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Obsessive Compulsive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Posttraumatic Stress | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Substance Abuse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Psychotic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Mood | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Anorexia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Bulemia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

| | Placebo | ANS-6637 300 mg | ANS-6637 600 mg | Total |
|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| Binge-eating | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Generalized Anxiety | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Medical Organic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Antisocial Personality | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

**Table 23:** Baseline POMS – mITT Subjects

| | Placebo | ANS-6637 200 | ANS-6637 600 mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| Characteristic | | mg | | | |
| Tension-Anxiety | | | | | 0.xxx |
| N | xx | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| $SD^2$ | xxx.xx | xxx.xx | XXX.XX | xxx.xx | |
| Median | xx | xx | XX | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |
| Depression-Dejection | | | | | 0.xxx |

| Characteristic | Placebo | ANS-6637 200<br>mg | ANS-6637 600 mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| N | XX | XX | xx | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XXX.XX | xxx.xx | xxx.xx | XXX.XX | |
| Median | XX | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |
| Anger-Hostility | | | | | 0.xxx |
| N | XX | XX | xx | XX | |
| Mean | XX.X | XX.X | xx.x | XX.X | |
| SD | XXX.XX | xxx.xx | xxx.xx | XXX.XX | |
| Median | XX | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |
| Fatigue-Inertia | | | | | 0.xxx |
| N | xx | XX | xx | XX | |
| Mean | xx.x | XX.X | xx.x | XX.X | |
| SD | XXX.XX | XXX.XX | xxx.xx | XXX.XX | |
| Characteristic | Placebo | ANS-6637 200<br>mg | ANS-6637 600 mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| onaracter istic | | •••• | | | |
| Median | xx | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |
| Confusion-Bewilderment | | | | | 0.xxx |
| N | xx | XX | xx | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | |
| Median | XX | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |
| Vigor-Activity | | | | | 0.xxx |
| N | xx | XX | xx | XX | |
| Mean | XX.X | XX.X | xx.x | XX.X | |
| SD | xxx.xx | XXX.XX | xxx.xx | XXX.XX | |
| Median | xx | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |

| Characteristic | Placebo | ANS-6637 200<br>mg | ANS-6637 600 mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| Total Mood Disturbance | | | | | 0.xxx |
| N | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | xxx.xx | XXX.XX | XXX.XX | XXX.XX | |
| Median | XX | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |

<sup>&</sup>lt;sup>1</sup>ANOVA F-test

**Table 24:** Baseline POMS – Evaluable Subjects

<sup>&</sup>lt;sup>2</sup>SD is standard deviation

**Table 25:** Baseline PSQI – mITT Subjects

| Characteristic | Placebo | ANS-6637 200 mg | ANS-6637 600 mg | Total | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| Overall Sleep Experience | | | | | 0.xxx |
| N | XX | XX | XX | XX | |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD <sup>2</sup> | xxx.xx | xxx.xx | XXX.XX | XXX.XX | |
| Median | XX | XX | xx | XX | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx-xx) | |

<sup>&</sup>lt;sup>1</sup>ANOVA F-test

 Table 26:
 Baseline PSQI – Evaluable Subjects

<sup>&</sup>lt;sup>2</sup> SD is standard deviation

 Table 27:
 Baseline Drinking-related Behavior and Characteristics – mITT Subjects

| | Placebo | ANS-6637 200 mg | ANS-6637 600 mg | Total | |
|---|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| Drinking Goal (n, %) | | | | | |
| Stop Drinking | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Reduce but not stop | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| # Drinks/Week Goal in Subjects tha | at Want to Reduce Drinking | | | | |
| N | xx | xx | XX | xx | 0.xxx |
| Mean | XX.X | XX.X | xx.x | xx.x | |
| SD <sup>2</sup> | xxx.xx | xxx.xx | xxx.xx | xxx.xx | |
| Median | XX | xx | XX | xx | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Motivation to achieve goal | | | | | |
| N | xx | xx | xx | xx | 0.xxx |
| Mean | XX.X | XX.X | XX.X | xx.x | |
| SD | xxx.xx | xxx.xx | xxx.xx | xxx.xx | |
| Median | xx | xx | xx | xx | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Confidence in achieving goal | | | | | |

| | Placebo | ANS-6637 200 mg | ANS-6637 600 mg | Total | |
|---|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| N | XX | xx | xx | xx | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX | |
| Median | xx | xx | xx | xx | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| AUD Symptom Severity (n, %) | | | | | 0.xxx |
| Moderate (4 or 5 symptoms) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Severe (6 or more symptoms) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| AUD Number of Symptoms (n, %) | | | | | |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 9 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 10 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| 11 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |

| | Placebo | ANS-6637 200 mg | ANS-6637 600 mg | Total | |
|---|---|---|---|---|---|
| Characteristic | (N=xx) | (N=xx) | (N=xx) | (N=xx) | p-value <sup>1</sup> |
| AUD Number of Symptoms (continuous) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | xx.x | |
| SD | XXX.XX | XXX.XX | xxx.xx | xxx.xx | |
| Median | XX | XX | XX | xx | |

Note: Percentages are based on the number of non-missing values in each variable.

 Table 28:
 Baseline Drinking-related Behavior and Characteristics – Evaluable Subjects

<sup>&</sup>lt;sup>1</sup> ANOVA F-test

<sup>&</sup>lt;sup>2</sup>SD is standard deviation

 Table 29:
 Baseline Drinking by TLFB – mITT Subjects

| | Placebo | ANS-6637<br>200mg | ANS-6637 600<br>mg | Total | |
|---|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Drinks/Week (Pre-screening Days -1 to -28) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD <sup>2</sup> | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Week (7 Days Prior to Randomization) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Week (Percent Change Pre-screening Days -1 to -28 to 7 Days Prior to Randomization) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |

| | Placebo | ANS-6637<br>200mg | ANS-6637 600<br>mg | Total | |
|---|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Drinks/Drinking Day (Pre-screening Days -1 to - 28) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Drinking Day (7Days Prior to<br>Randomization) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Drinks/Drinking Day (Percent Change Prescreening Days -1 to -28 to 7 Days Prior to Randomization) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |

| | Placebo | ANS-6637<br>200mg | ANS-6637 600<br>mg | Total | |
|---|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Percentage of Heavy Drinking Days<br>(Pre-screening Days -1 to -28) | | | | | 0.xxx |
| Mean | xx.x% | xx.x% | xx.x% | xx.x% | |
| SD | xx.x% | xx.x% | xx.x% | xx.x% | |
| Median | xx.x% | xx.x% | xx.x% | xx.x% | |
| Min-Max | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | |
| Percentage of Very Heavy Drinking Days<br>(Pre-screening Days -1 to -28) | | | | | 0.xxx |
| Mean | xx.x% | xx.x% | xx.x% | xx.x% | |
| SD | xx.x% | xx.x% | xx.x% | xx.x% | |
| Median | xx.x% | xx.x% | xx.x% | xx.x% | |
| Min-Max | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | |
| Percentage Days Abstinent<br>(Pre-screening Days -1 to -28) | | | | | 0.xxx |
| Mean | xx.x% | xx.x% | xx.x% | xx.x% | |
| SD | xx.x% | xx.x% | xx.x% | xx.x% | |

| | Placebo | ANS-6637 | ANS-6637 600 | Total | |
|---|---|---|---|---|---|
| | | 200mg | mg | | |
| Parameter | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Median | xx.x% | xx.x% | xx.x% | xx.x% | |
| Min-Max | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | (xx%-xx%) | |
| WHO Risk Level | | | | | 0.xxx |
| High Risk | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Very High Risk | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Note: Percentages are based on the number of non-missing values in each variable.

**Table 30:** Baseline Drinking by TLFB – Evaluable Subjects

<sup>&</sup>lt;sup>1</sup>Chi-square test for categorical variables and ANOVA F-test for continuous variables

<sup>&</sup>lt;sup>2</sup> SD is standard deviation

Table 31: Baseline Alcohol-Related Craving, Consequences, Withdrawal and ALDH2 – mITT Subjects

Placebo ANS-6637 ANS-6637 600 **Total** mg 200mg p-value<sup>1</sup> **Parameter** (N=xx)(N=xx)(N=xx)(N=xxx)Pre-cue ACQ-SF-R<sup>2</sup> 0.xxxMean XX.X XX.X XX.X XX.X SD<sup>3</sup> XX.X XX.X XX.X XX.X Median XX.X XX.X XX.X XX.X Min-Max (xx-xx) (xx-xx) (xx-xx) (xx-xx) Scale Min-Max (xx.x - xx.x)Post-cue ACQ-SF-R 0.xxx Mean XX.X XX.X XX.X XX.X SD XX.X XX.X XX.X XX.X Median XX.X XX.X XX.X XX.X Min-Max (xx-xx) (xx-xx) (xx-xx)(xx-xx)Pre-Post ACQ-SF-R Mean XX.X XX.X XX.X XX.X SD XX.X XX.X XX.X XX.X Median XX.X XX.X XX.X XX.X

| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
|---|---|---|---|---|---|
| PROMIS <sup>4</sup> Alcohol Negative<br>Consequences (T-scores) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| PACS <sup>5</sup> | | | | | 0.xxx |
| Mean | XX.X | xx.x | XX.X | XX.X | |
| SD | XX.X | xx.x | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Scale Min-Max | | | | (xx.x - xx.x) | |
| CIWA-AR <sup>6</sup> | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Maximum | XX.X | XX.X | XX.X | XX.X | |

| | Placebo | ANS-6637<br>200mg | ANS-6637 600<br>mg | Total | |
|---|---|---|---|---|---|
| Parameter | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Scale Min-Max | | | | (xx.x - xx.x) | |
| Withdrawal Symptoms (CIWA ≥ 10) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| ALDH2 | | | | | 0.xxx |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Not Done | XX | XX | XX | XX | |

<sup>&</sup>lt;sup>1</sup>ANOVA F-test for continuous variables and chi-square test for categorical

**Table 32:** Baseline Alcohol-Related Craving, Consequences, Withdrawal and ALDH2 – Evaluable Subjects

Same as Table 31

<sup>&</sup>lt;sup>2</sup>ACQ-SF-R is Alcohol Craving Questionnaire – Short Form – Revised

<sup>&</sup>lt;sup>3</sup> SD is standard deviation

<sup>&</sup>lt;sup>4</sup> PROMIS is Patient-reported Outcomes Information System

<sup>&</sup>lt;sup>5</sup> PACS is Penn Alcohol Craving Scale

<sup>&</sup>lt;sup>6</sup> CIWA-AR is Clinical Institute Withdrawal Assessment for Alcohol-revised

 Table 33:
 Baseline Other Substance Use – mITT Subjects

| | Placebo | ANS-6637 | ANS-6637 600 mg | Total | |
|---|---|---|---|---|---|
| | | 200 mg | | | |
| Parameter | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| Smoker (n, %) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | 0.xxx |
| Days Smoked in the Past Week | | | | | |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD <sup>2</sup> | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| (Min-Max) | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Average Cigarettes Smoked Per Week (among Smokers) | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | XX.X | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Any Other Nicotine Product Use (doesn't include cigarettes) (n, %) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | 0.xxx |
| Days Used Other Nicotine Products Per Week | | | | | 0.xxx |
| Mean | XX.X | XX.X | XX.X | XX.X | |

| | Placebo | ANS-6637 | ANS-6637 600 mg | Total | |
|---|---|---|---|---|---|
| | | 200 mg | | | |
| Parameter | (N=xx) | (N=xx) | (N=xx) | (N=xxx) | p-value <sup>1</sup> |
| SD | XX.X | XX.X | XX.X | XX.X | |
| Median | XX.X | xx.x | XX.X | XX.X | |
| Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) | |
| Any Nicotine Use (cigarettes + other) (n, %) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | 0.xxx |
| ТНС | | | | | 0.xxx |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Positive | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

Note: Percentages are based on the number of non-missing values in each variable.

**Table 34:** Baseline Other Substance Use – Evaluable Subjects

<sup>&</sup>lt;sup>1</sup>ANOVA F-test for continuous variables and chi-square test for categorical

<sup>&</sup>lt;sup>2</sup> SD is standard Deviation

# 12.1.3. Primary Efficacy Endpoint

 Table 35:
 Week 2 Strength of Craving Scores – mITT Subjects

| | | Placebo | ANS-6637 200 mg | ANS-6637 | Total |
|---|---|---|---|---|---|
| | | N=xx | N=xx | 600 mg | N=xx |
| | | | | N=xx | |
| Cue | Statistic | | | | |
| Water | | | | | |
| | Mean (SD <sup>1</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | xx | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 1 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | xx | XX | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | xx | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 1 - Water | | | | | |

| | | Placebo<br>N=xx | ANS-6637 200 mg<br>N=xx | ANS-6637<br>600 mg<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | xx | xx | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 - Water | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | xx | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 –<br>Alcohol 1 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | xx | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

Week 2 Strength of Craving<sup>1</sup> Scores – Evaluable Subjects **Table 36:** 

Same as Table 35

Table 37: ANCOVA Strength of Craving<sup>1</sup> – mITT Subjects

Type III Wald Tests

| Parameter | Num DF <sup>2</sup> | Den DF <sup>3</sup> | F Value | p-value |
|---|---|---|---|---|
| ARM | 2 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>4</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Strength of craving from 1<sup>st</sup> alcohol cue; <sup>32</sup>Numerator degrees of freedom; <sup>3</sup> Demonimator degrees of freedom

| Arm | Mean | SE <sup>1</sup> | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
|---|---|---|---|---|---|
| placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 200 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test; <sup>3</sup> Lower and upper limit of 95% confidence interval

<sup>&</sup>lt;sup>4</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

## **Least Squares Means for Differences**

| | | | | | | Tukey | |
|---|---|---|---|---|---|---|---|
| Arm1 | Arm 2 | Difference | SE <sup>1</sup> | Cohen's d | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
| 200 mg | placebo | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | placebo | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | 200 mg | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Tukey's test; <sup>3</sup> Lower and upper limit of 95% confidence interval

Table 38: ANCOVA Strength of Craving – Evaluable Subjects

Follow the same analysis as Table 37

| 12.1.4. | . Confirmatory Secondary Efficacy Endpoints |
|---------|---------------------------------------------|

Table 39: ANCOVA Strength of Craving (Difference Alcohol-Water) – mITT Subjects

Type III Wald Test

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| ARM | 2 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>4</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup>Strength of craving from 1<sup>st</sup> alcohol cue; <sup>2</sup>Numerator degrees of freedom; <sup>3</sup> Demonimator degrees of freedom

### **Least Squares Means Difference**

| | | | | | | Tukey | |
|---|---|---|---|---|---|---|---|
| Arm1 | Arm 2 | Difference | $SE^1$ | Cohen's d | p-value <sup>2</sup> | Lower CI <sup>1</sup> | Upper CI |
| 200 mg | placebo | xx.xx | 0.xxx | x.xx | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | placebo | xx.xx | 0.xxx | x.xx | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | 200 mg | xx.xx | 0.xxx | x.xx | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Tukey's test; <sup>3</sup> Lower and upper limit of 95% confidence interval

| Arm | Mean | SE <sup>1</sup> | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

<sup>&</sup>lt;sup>4</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

| Arm | Mean | SE <sup>1</sup> | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
|---|---|---|---|---|---|
| placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 200 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test; <sup>3</sup> Lower and upper limit of 95% confidence interval

**Table 40:** ANCOVA Strength of Craving (Difference Alcohol-Water) – Evaluable Subjects Same as Table 39

**Table 41:** Drinking Makes Things Perfect Scores – mITT Subjects

| | | Placebo<br>N=xx | ANS-6637 200<br>mg<br>N=xx | ANS-6637<br>600 mg<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Cue | Statistic | | | | |
| Water | | | | | |
| | Mean (SD <sup>1</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | XX | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 1 | | | | | |

| | | Placebo<br>N=xx | ANS-6637 200<br>mg<br>N=xx | ANS-6637<br>600 mg<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | XX | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 1 - Water | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 - Water | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |

| | | Placebo<br>N=xx | ANS-6637 200<br>mg<br>N=xx | ANS-6637<br>600 mg<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Alcohol 2 –<br>Alcohol 1 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | XX | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

**Table 42:** Drinking Makes Things Perfect Scores – Evaluable Subjects

Table 43: ANCOVA Drinking Makes Things Perfect<sup>1</sup> – mITT Subjects

Type III Wald Test

| Parameter | Num DF <sup>2</sup> | Den DF <sup>3</sup> | F Value | p-value |
|---|---|---|---|---|
| ARM | 2 | XX | xxx.xx | 0.xxx |
| Site | 2 | XX | xxx.xx | 0.xxx |
| Baseline Cue <sup>4</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Drinking makes things perfect from 1<sup>st</sup> alcohol cue; <sup>2</sup>Numerator degrees of freedom; <sup>3</sup> Demonimator degrees of freedom

| Arm | Mean | SE <sup>1</sup> | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
|---|---|---|---|---|---|
| placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 200 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test; <sup>3</sup> Lower and upper limit of 95% confidence interval

<sup>&</sup>lt;sup>4</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

# **Least Squares Means for Differences**

| | | | | | | Tukey | |
|---|---|---|---|---|---|---|---|
| Arm1 | Arm 2 | Difference | $SE^1$ | Cohen's d | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
| 200 mg | placebo | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | placebo | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | 200 mg | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |

 $<sup>^1</sup>$  SE is standard error;  $^2$  Tukey's test;  $^3$  Lower and upper limit of 95% confidence interval

Table 44: ANCOVA Drinking Makes Things Perfect – Evaluable Subjects

Table 45: ANCOVA Drinking Makes Things Perfect<sup>1</sup> (Difference Alcohol-Water) – mITT Subjects

Type III Wald Test

| Parameter | Num DF <sup>2</sup> | Den DF <sup>3</sup> | F Value | p-value |
|---|---|---|---|---|
| ARM | 2 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>4</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Drinking makes things perfect from 1<sup>st</sup> alcohol cue; <sup>2</sup>Numerator degrees of freedom; <sup>3</sup> Demonimator degrees of freedom

#### **Least Squares Means Differences**

| | | | | | | Tukey | |
|---|---|---|---|---|---|---|---|
| Arm1 | Arm 2 | Difference | SE <sup>1</sup> | Cohen's d | p-value <sup>2</sup> | Lower CI <sup>1</sup> | Upper CI |
| 200 mg | placebo | xx.xx | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | placebo | xx.xx | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | 200 mg | xx.xx | 0.xxx | x.xx | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Tukey's test; <sup>3</sup> Lower and upper limit of 95% confidence interval

<sup>&</sup>lt;sup>4</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

**Least Squares Means** 

| Arm | Mean | SE <sup>1</sup> | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
|---|---|---|---|---|---|
| placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 200 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test; <sup>3</sup> Lower and upper limit of 95% confidence interval

**Table 46:** ANCOVA Drinking Makes Things Perfect (Difference Alcohol-Water) – Evaluable Subjects Same analysis as Table 45

Table 47: Drink Now Scores- mITT Subjects

| | | Placebo<br>N=xx | ANS-6637 200<br>mg<br>N=xx | ANS-6637<br>600 mg<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| Cue | Statistic | | | | |
| Water | | | | | |
| | Mean (SD <sup>1</sup> ) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 1 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | xx | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 1 - Water | | | | | |

| | | Placebo<br>N=xx | ANS-6637 200<br>mg<br>N=xx | ANS-6637<br>600 mg<br>N=xx | Total<br>N=xx |
|---|---|---|---|---|---|
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 - Water | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx | XX | XX | XX |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |
| Alcohol 2 –<br>Alcohol 1 | | | | | |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX | XX | xx | xx |
| | Min-Max | (xx-xx) | (xx-xx) | (xx-xx) | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

 Table 48:
 Drink Now Scores – Evaluable Subjects

**Table 49:** ANCOVA Drink Now<sup>1</sup> – mITT Subjects

**Type III Wald Test** 

| Parameter | Num DF <sup>2</sup> | Den DF <sup>3</sup> | F Value | p-value |
|---|---|---|---|---|
| ARM | 2 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| Baseline Cue <sup>4</sup> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Drinking now from 1<sup>st</sup> alcohol cue; <sup>2</sup>Numerator degrees of freedom; <sup>3</sup> Demonimator degrees of freedom

| Arm | Mean | SE <sup>1</sup> | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
|---|---|---|---|---|---|
| placebo | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 200 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | XX.XX | 0.xxx | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Wald test; <sup>3</sup> Lower and upper limit of 95% confidence interval

<sup>&</sup>lt;sup>4</sup> Baseline Cue is the baseline equivalent of the outcome obtained after the presentation of the first alcohol cue at baseline

### **Least Squares Means for Differences**

| | | | | | | Tukey | |
|---|---|---|---|---|---|---|---|
| Arm1 | Arm 2 | Difference | $SE^1$ | Cohen's d | p-value <sup>2</sup> | Lower CI <sup>3</sup> | Upper CI |
| 200 mg | placebo | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | placebo | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |
| 600 mg | 200 mg | XX.XX | 0.xxx | X.XX | 0.xxx | 0.xxx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> Tukey's test; <sup>3</sup> Lower and upper limit of 95% confidence interval

**Table 50:** ANCOVA Drink Now<sup>1</sup> – Evaluable Subjects

Same analysis as Table 49

Table 51: ANCOVA Drink Now<sup>1</sup> (Difference Alcohol-Water) – mITT Subjects

Same analysis as Table 45 with difference as the dependent variable

Table 52: ANCOVA Drink Now<sup>1</sup> (Difference Alcohol-Water) – Evaluable Subjects

Same analysis as Table 51

**Table 53:** Turn Down Drink Scores – mITT Subjects

Same analysis as Table 47

**Table 54:** Turn Down Drink Scores – Evaluable Subjects

**Table 55:** ANCOVA Turn Down Drink<sup>1</sup> – mITT Subjects

Same analysis as Table 49

**Table 56:** ANCOVA Turn Down Drink<sup>1</sup> – Evaluable Subjects

Same analysis as Table 55

Table 57: ANCOVA Turn Down Drink<sup>1</sup> (Difference Alcohol-Water) – mITT Subjects

Same analysis as Table 45

Table 58: ANCOVA Turn Down Drink<sup>1</sup> (Difference Alcohol-Water) – Evaluable Subjects

Same analysis as Table 57

**Table 59:** Average of Cue Scores – mITT Subjects

Same analysis as Table 47

**Table 60:** Average of Cue Scores – Evaluable Subjects

Same as Table 59

Table 61: ANCOVA Average of Cue Scores<sup>1</sup> – mITT Subjects

Same analysis as Table 49

Table 62: ANCOVA Average of Cue Scores<sup>1</sup> – Evaluable Subjects

Same analysis as Table 61

Table 63: ANCOVA Average of Cue Scores<sup>1</sup> (Difference Alcohol-Water) – mITT Subjects

Same analysis as Table 45

Table 64: ANCOVA Average of Cue Scores<sup>1</sup> (Difference Alcohol-Water) – Evaluable Subjects

**Table 65:** Beverage Liking Scores – mITT Subjects

Same analysis as Table 47

**Table 66:** Beverage Liking Scores – Evaluable Subjects

| 12.1.5. | <b>Secondary</b> | <b>Efficacy</b> | <b>Endpoints</b> |
|---------|------------------|-----------------|------------------|
Table 67: Percentage of Subjects No Heavy Drinking Days Weeks 2-5 – mITT Subjects

| | | <b>ANS-6637</b> | ANS-6637 | |
|---|---|---|---|---|
| | Placebo | 200 mg | 600 mg | Total |
| | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| No Heavy Drinking Days | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 68: Percentage of Subjects with No Heavy Drinking Days Weeks 2-5 – Full Model Logistic Regression (mITT)

| | | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | $\mathbf{DF}^1$ | Estimate | Standard | Wald | Pr > Chi- | Cohen's h | $OR^2$ | Upper CI | Lower CI |
| | | | | Error | Chi-Square | Square | | | | |
| Intercept | | 1 | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment <sup>4</sup> | 200 mg | X | XX.XXX | XX.XXX | xx.xxx | 0.xxx | 0.xxx | xx.xxx | xx.xxx | XX.XXX |
| Treatment | 600 mg | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | 0.xxx | xx.xxx | xx.xxx | XX.XXX |
| Site | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |

| | | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF <sup>1</sup> | Estimate | Standard<br>Error | Wald<br>Chi-Square | | Cohen's h | OR <sup>2</sup> | Upper CI | Lower CI |
| Site <sup>5</sup> | 1 | X | XX.XXX | XX.XXX | xx.xxx | 0.xxx | | xx.xxx | xx.xxx | xx.xxx |
| Site | 2 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | xx.xxx | xx.xxx | xx.xxx |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | XX.XXX | xx.xxx | xx.xxx |

<sup>&</sup>lt;sup>1</sup> DF is degrees of freedom; <sup>2</sup> OR is odds ratio; <sup>3</sup> CI is confidence interval; <sup>4</sup> Comparison to placebo for each active treatment;

Programming note: COV is baseline equivalent of dependent variable and any other covariate(s) which have not been specified at the time of writing of SAP

#### Contrast

| | | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | $\mathbf{DF}^1$ | Estimate | | | Pr > Chi- Cohen's h | | $OR^2$ | Upper CI | Lower CI |
| | | | | Error | Chi-Square | Square | | | | |
| 600 mg | 200 mg | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | 0.xxx | XX.XXX | xx.xxx | xx.xxx |

<sup>&</sup>lt;sup>1</sup> DF is degrees of freedom; <sup>2</sup> OR is odds ratio; <sup>3</sup> CI is confidence interval.

## Table 69: Percentage of Subjects Abstinent from Alcohol Weeks 2-5 – mITT Subjects

Presented in same manner as Table 67

<sup>&</sup>lt;sup>5</sup> Site 3 is reference for the OR

Table 70: Percentage of Subjects Abstinent from Alcohol Weeks 2-5 – Full Model Logistic Regression (mITT)

Prented in same manner as Table 68 programming note: baseline PDA is a covariate for PSA outcome

Table 71: WHO 1-Level Decrease in Alcohol Consumption (mITT) – Weeks 2-5

| | Placebo | ANS-6637<br>200mg | ANS-6637<br>600 mg | Total |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| WHO 1-Level<br>Decrease | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 72: WHO 1-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 2-5

| | | | | | | | | | 95% | CI <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF <sup>1</sup> | Estimate | Standard<br>Error | Wald Chi-<br>Square | Pr > Chi-<br>Square | Cohen's<br>h | $OR^2$ | Upper CI | Lower CI |
| Intercept | | 1 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment | Overall | 2 | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Treatment <sup>4</sup> | 200mg | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | 0.xxx | XX.XXX | XX.XXX | XX.XXX |
| Treatment | 600mg | Х | xx.xxx | XX.XXX | XX.XXX | 0.xxx | 0.xxx | xx.xxx | XX.XXX | XX.XXX |
| Site | Overall | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | | | |
| Site <sup>5</sup> | 1 | Х | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | XX.XXX | XX.XXX |
| Site | 2 | Х | xx.xxx | xx.xxx | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |
| Cov | | X | XX.XXX | XX.XXX | XX.XXX | 0.xxx | | xx.xxx | XX.XXX | XX.XXX |

<sup>&</sup>lt;sup>1</sup> DF is degrees of freedom; <sup>2</sup> OR is odds ratio; <sup>3</sup> CI is confidence interval; <sup>4</sup> Comparison to placebo for each active treatment;

Programming note: COV is baseline equivalent of dependent variable and any other covariate(s) which have not been specified at the time of writing of SAP

#### Contrast

| | | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Param | ieter | DF <sup>1</sup> | Estimate | Standard<br>Error | Wald<br>Chi-Square | | Cohen's h | OR <sup>2</sup> | Upper CI | Lower CI |
| 600 mg | 200 mg | 1 | XX.XXX | XX.XXX | xx.xxx | 0.xxx | 0.xxx | xx.xxx | xx.xxx | xx.xxx |

<sup>&</sup>lt;sup>1</sup> DF is degrees of freedom; <sup>2</sup> OR is odds ratio; <sup>3</sup> CI is confidence interval.

<sup>&</sup>lt;sup>5</sup> Site 3 is reference for the OR

Table 73: WHO 2-Level Decrease in Alcohol Consumption (mITT) – Weeks 2-5

Same as Table 71

Table 74: WHO 2-Level Decrease in Alcohol Consumption (mITT) – Full Model, Logistic Regression, Weeks 2-5

Same as Table 72

Table 75: Percentage of Days Abstinent per Week (mITT) – Weeks 2-5

| | | | | | | ANS-6637 | • | | | ANS-6637 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Placebo | | | | 200mg | | | 600 mg | | | |
| Study<br>Week | N | Mean (SD¹) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |
| 2 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | xxx | (xx-xx) | XX | xxx (xx) | xxx | (xx-xx) |
| 3 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 4 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 5 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |

SD is standard deviation

Table 76: Percentage of Days Abstinent per Week (mITT) -- Full Model, Mixed Effects, Weeks 2-5

Type III Wald Tests

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|-----------|---------------------|---------------------|---------|---------|
| ARM | 2 | xxx | xxx.xx | 0.xxx |
| Week | 3 | XXX | XXX.XX | 0.xxx |
| Site | 2 | XXX | XXX.XX | 0.xxx |
| Cov | Х | XXX | XXX.XX | 0.xxx |
| ARM*Week | 5 | XXX | XXX.XX | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Numerator degrees of freedom; <sup>2</sup> Denominator degrees of freedom

Programming note: Cov is the baseline equivalent of the dependent variable and any additional covariates included in the model.

# **Least Squares Means**

| | | | | 95% CI <sup>2</sup> | | | | | sformed |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(200mg) | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 2 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |
| ANS-6637<br>(200mg) | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

| | | | | 959 | % CI <sup>2</sup> | | | Untran | sformed |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(200mg) | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| ANS-6637<br>(200mg) | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| ANS-6637<br>(200mg) | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

#### **Contrasts**

| | | | | 95% CI <sup>3</sup> | | | | | Untransformed |
|---|---|---|---|---|---|---|---|---|---|
| Arm <sup>1</sup> | Week | Estimate | SE <sup>2</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(600mg) | 2 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 3 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |

| | | | | 95% | % CI <sup>3</sup> | | | Untransformed | |
|---|---|---|---|---|---|---|---|---|---|
| Arm <sup>1</sup> | Week | Estimate | SE <sup>2</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(600mg) | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 5 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |

 $<sup>^{1}</sup>$  ANS-6637 200 mg is the reference group;  $^{2}$  SE is standard error;  $^{3}$  CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

Table 75 is the template for Tables 77, 79, 81, 83, 85, and 87. Table 76 is the template for Tables 78, 80, 82, 84, 86, and 88.

Table 77: Percentage of Heavy Drinking Days per Week (mITT) – Weeks 2-5

Table 78: Percentage of Heavy Drinking Days per Week (mITT) – Full Model, Mixed Effects, Weeks 2-5

Table 79: Percentage of Very Heavy Drinking Days per Week (mITT) – Weeks 2-5

Table 80: Percentage of Very Heavy Drinking Days per Week (mITT) – Full Model, Mixed Effects, Weeks 2-5

Table 81: Drinks per Week (mITT) – Weeks 2-5

Table 82: Drinks per Week (mITT) – Full Model, Mixed Effects, Weeks 2-5

Table 83: Drinks per Drinking Day (mITT) – Weeks 2-5

Table 84: Drinks per Drinking Day (mITT) – Full Model, Mixed Effects, Weeks 2-5

Table 85: Mean Cigarettes Smoked Among Smokers (mITT) – Weeks 2-5

Table 86: Mean Cigarettes Smoked Among Smokers (mITT) – Full Model, Mixed Effects, Weeks 2-5

Table 87: PACS (mITT) – Weeks 2-5

Table 88: PACS (mITT) – Full Model, Mixed Effects, Weeks 2-5

Table 89: Percentage of Subjects Abstinent from Nicotine Use<sup>1</sup> Weeks 2-5 – Among Subjects that Used Nicotine Products at Baseline

| | Placebo | ANS-6637<br>200 mg | ANS-6637 600<br>mg | Total |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| No Nicotine Use | | | | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

<sup>&</sup>lt;sup>1</sup> Nicotine use includes cigarettes or other nicotine products

Table 90: Percentage of Subjects Abstinent from Nicotine Use<sup>1</sup> Weeks 2-5 – Full Model Logistic Regression (Among Nicotine Users at Baseline)

| | | | | | | | | | 95% CI <sup>4</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | $\underset{2}{\mathbf{DF}}$ | Estimate | Standard | Wald | | Cohen's h | OR <sup>3</sup> | Upper CI | Lower CI |
| | | , | | Error | Chi-Square | Square | 1 | | | |
| Intercept | | 1 | xx.xxx | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Treatment <sup>5</sup> | 200 mg | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | 0.xxx | XX.XXX | xx.xxx | xx.xxx |
| Treatment | 600 mg | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | 0.xxx | XX.XXX | xx.xxx | xx.xxx |

| | | | | | | | | | 95% CI <sup>4</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | | DF | Estimate | Standard | Wald | Pr > Chi- | Cohen's h | $OR^3$ | Upper CI | Lower CI |
| | | 2 | | Error | Chi-Square | Square | | | | |
| Site | Overall | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | | | |
| Site <sup>6</sup> | 1 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | xx.xxx | XX.XXX |
| Site | 2 | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | xx.xxx | XX.XXX |
| Cov | | X | XX.XXX | xx.xxx | xx.xxx | 0.xxx | | XX.XXX | xx.xxx | xx.xxx |

<sup>&</sup>lt;sup>1</sup> Nicotine use includes either cigarettes or other nicotine products; <sup>2</sup> DF is degrees of freedom; <sup>3</sup> OR is odds ratio; <sup>4</sup> CI is confidence interval; <sup>5</sup> Comparison to placebo for each active treatment; <sup>6</sup> Site 3 is reference for the OR

Programming note: COV is baseline equivalent of dependent variable and any other covariate(s) which have not been specified at the time of writing of SAP

#### Contrast

| | | | | | | | | | 95% CI <sup>3</sup> | |
|---|---|---|---|---|---|---|---|---|---|---|
| Param | eter | DF <sup>1</sup> | Estimate | Standard<br>Error | Wald<br>Chi-Square | | Cohen's h | OR <sup>2</sup> | Upper CI | Lower CI |
| 600 mg | 200 mg | 1 | XX.XXX | XX.XXX | xx.xxx | 0.xxx | 0.xxx | xx.xxx | xx.xxx | XX.XXX |

<sup>&</sup>lt;sup>1</sup> DF is degrees of freedom; <sup>2</sup> OR is odds ratio; <sup>3</sup> CI is confidence interval.

Table 91: Percentage of Subjects Abstinent from Smoking Weeks 2-5 – Among Baseline Smokers

Same analysis as Table 89

Table 92: Percentage of Subjects Abstinent from Smoking Weeks 2-5 – Full Model Logistic Regression (Among Baseline Smokers)

Same analysis as Table 90

**Table 93:** PSQI Scores – mITT Subjects

| | | | | | | ANS-6637 | , | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Placebo 200mg | | | | | | | 600 mg | | | |
| Study | | | | | | | | | | | | |
| Week | N | Mean (SD¹) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

**Table 94:** ANCOVA PSQI Score – mITT Subjects

**Type III Wald Tests** 

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| ARM | 2 | xx | XXX.XX | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| <b>Baseline PSQI</b> | 1 | xx | XXX.XX | 0.xxx |

# **Least Squares Means**

| | | | | 95% CI <sup>2</sup> | | | | Untransformed | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower<br>CI | Upper CI | I Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(200mg) | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | X.XXX | 0.xxx | xx.xxx |
| Placebo | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

#### **Contrasts**

| | | | | 95% CI <sup>3</sup> | | | | | Untransformed |
|---|---|---|---|---|---|---|---|---|---|
| Arm <sup>1</sup> | Week | Estimate | SE <sup>2</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(600mg) | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |

 $<sup>^{1}</sup>$  ANS-6637 200 mg is the reference group;  $^{2}$  SE is standard error;  $^{3}$  CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

**Table 95: POMS Total Mood Disturbance Score – mITT** 

| | | TOMS I | 7tai 14100u | Distui Dance | Score | ANS-6637 | , | | ANS-6637 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Placebo 200mg | | | | | | | 600 mg | | | | |
| Study<br>Week | N | Mean (SD¹) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |
| 4 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |
| 6 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

Table 96: POMS Total Mood Disturbance Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6

Type III Wald Tests

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|-----------|---------------------|---------------------|---------|---------|
| ARM | 2 | xxx | xxx.xx | 0.xxx |
| Week | 1 | xxx | xxx.xx | 0.xxx |
| Site | 2 | xxx | xxx.xx | 0.xxx |
| Cov | X | xxx | xxx.xx | 0.xxx |
| ARM*Week | X | xxx | xxx.xx | 0.xxx |

# <sup>1</sup> Numerator degrees of freedom; <sup>2</sup> Denominator degrees of freedom

Programming note: Cov is the baseline equivalent of the dependent variable and any additional covariates included in the model.

# **Least Squares Means**

| | | | | 95% CI <sup>2</sup> | | | | Untransfo | rmed |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(200mg) | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| ANS-6637<br>(200mg) | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |
| ANS-6637<br>(200mg) | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| Placebo | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

## **Contrasts**

| | | | | 95% CI <sup>3</sup> | | | | Untransformed | |
|---|---|---|---|---|---|---|---|---|---|
| Arm <sup>1</sup> | Week | Estimate | SE <sup>2</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(600mg) | 4 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |
| ANS-6637<br>(600mg) | Overall | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |

 $<sup>^{1}</sup>$  ANS-6637 200 mg is the reference group;  $^{2}$  SE is standard error;  $^{3}$  CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

Table 95 is the template for Tables 97, 99, 101, 103, 105, and 107. Table 96 is the template for Tables 98, 100, 102, 104, 106, and 108

**Table 97:** POMS Tension-Anxiety Score – mITT Subjects

Table 98: POMS Tension-Anxiety Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6

**Table 99:** POMS Anger-Hostility Score – mITT Subjects

Table 100: POMS Anger-Hostility Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6

**Table 101: POMS Vigor-Activity Score – mITT Subjects** 

Table 102: POMS Vigor-Activity Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6

**Table 103:** POMS Fatigue-Inertia Score – mITT Subjects

Table 104: POMS Fatigue-Inertia Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6

**Table 105 POMS Confusion-Bewilderment Score – mITT Subjects** 

Table 106: POMS Confusion-Bewilderment Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6

**Table 107:** POMS Depression-Dejection Score – mITT Subjects

Table 108: POMS Depression-Dejection Score (mITT) – Full Model, Mixed Effects, Weeks 4 + 6

**Table 109:** PROMIS Negative Consequences of Alcohol Scores – mITT Subjects

| | | | | | ANS-6637 | | | ANS-6637 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | F | Placebo | | 200mg 600 mg | | | | | | | |
| Study<br>Week | N | Mean (SD¹) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) | N | Mean (SD) | Median | (Min-Max) |
| 6 | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) | XX | xxx (xx) | XXX | (xx-xx) |

<sup>&</sup>lt;sup>1</sup> SD is standard deviation

Table 110: ANCOVA PROMIS Negative Consequences of Alcohol – mITT Subjects

Type III Wald Test

| Parameter | Num DF <sup>1</sup> | Den DF <sup>2</sup> | F Value | p-value |
|---|---|---|---|---|
| ARM | 2 | xx | xxx.xx | 0.xxx |
| Site | 2 | xx | xxx.xx | 0.xxx |
| <b>Baseline PROMIS</b> | 1 | xx | xxx.xx | 0.xxx |

<sup>&</sup>lt;sup>1</sup> Numerator degrees of freedom; <sup>2</sup> Demonimator degrees of freedom

# **Least Squares Means**

| | | | | 95% CI <sup>2</sup> | | | | Untransformed | |
|---|---|---|---|---|---|---|---|---|---|
| Arm | Week | Estimate | SE <sup>1</sup> | Lower<br>CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637 (200mg) | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | X.XXX | 0.xxx | xx.xxx |
| ANS-6637 (600mg) | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | X.XXX | x.xxx | 0.xxx | xx.xxx |
| Placebo | 6 | XX.XX | 0.xxx | 0.xxx | 0.xxx | | | | |

<sup>&</sup>lt;sup>1</sup> SE is standard error; <sup>2</sup> CI is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

# Contrasts

| | | | | 95% CI <sup>3</sup> | | | | Untransformed | |
|---|---|---|---|---|---|---|---|---|---|
| Arm <sup>1</sup> | Week | Estimate | SE <sup>2</sup> | Lower CI | Upper CI | Difference | SE | p-value | Cohen's d |
| ANS-6637<br>(600mg) | 6 | xx.xx | 0.xxx | 0.xxx | 0.xxx | x.xxx | x.xxx | 0.xxx | xx.xxx |

 $<sup>^{1}</sup>$  ANS-6637 200 mg is the reference group;  $^{2}\,\mathrm{SE}$  is standard error;  $^{3}\,\mathrm{CI}$  is confidence interval

Programming note: If a transformation of the dependent variable is used add 2 columns: p-value and Cohen's d for the transformed model.

# 12.1.6. Safety Analyses

 Table 111:
 Overall Summary of Adverse Events – Safety Subjects

| | Placebo | ANS-6637-<br>200mg | ANS-6637 600<br>mg | Total |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| Number of AEs | xx | XX | xx | XX |
| Number of SAEs | XX | XX | XX | XX |
| Number (%) of subjects with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number (%) of subjects with at least one SAE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number (%) of subjects with at least one AE related <sup>1</sup> to study product | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Number of AEs by severity | | | | |
| Mild | XX | XX | XX | XX |
| Moderate | XX | XX | XX | XX |
| Severe | XX | XX | XX | XX |
| Number of AEs by relationship to study product | | | | |
| At least possibly related | XX | XX | XX | XX |
| Unrelated | XX | XX | XX | XX |
| Number of AEs by SAE status | | | | |

| | Placebo | ANS-6637-<br>200mg | ANS-6637 600<br>mg | Total |
|-----|---------|--------------------|--------------------|---------|
| | (N=xx) | (N=xx) | (N=xx) | (N=xxx) |
| No | XX | XX | XX | XX |
| Yes | XX | XX | XX | XX |

<sup>&</sup>lt;sup>1</sup> Related is possible, probable, or definite

**Table 112:** Overall Summary of Adverse Events p-values – Safety Subjects

| | o verum summary of fluverse Events p values | ANS-6637 200<br>mg vs Placebo | ANS-6637 600<br>mg vs Placebo | ANS-6637 200 mg vs<br>ANS-6637 600 mg |
|---|---|---|---|---|
| Number of s | subjects with at least one AE | 0.xxx | 0.xxx | 0.xxx |
| Number of s | subjects with at least one SAE | 0.xxx | 0.xxx | 0.xxx |
| Number of s | subjects with at least one AE related to study product | 0.xxx | 0.xxx | 0.xxx |

p-value from chi-square test (c), unless a row has expected fewer than 5 in a cell then Fisher's exact test (f)

Table 113: Number and Percentage of Subjects with Adverse Events - Safety Subjects

| MedDRA System Organ Class/ | Placebo | ANS-6637-200mg | ANS-6637 600 mg |
|----------------------------|------------|----------------|-----------------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| - Any Adverse Events - | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SOC | | | |
| - Overall - | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 114: Number and Percentage of Subjects with Adverse Events p-values - Safety Subjects

| MedDRA System Organ Class | ANS-6637 200 mg<br>vs Placebo | ANS-6637 600 mg<br>vs Placebo | ANS-6637 200 mg<br>vs ANS-6637 600<br>mg |
|---|---|---|---|
| Gastrointestinal disorders | 0.xxx | 0.xxx | 0.xxx |
| Infections and infestations | 0.xxx | 0.xxx | 0.xxx |

p-value from chi-square test (c), unless a row has expected fewer than 5 in a cell then Fisher's exact test (f)

Programming note: Include all SOCs that are in Table 111

Statistical Analysis Plan: Protocol HLAB-002, Version 1.0 Dated: 16Mar2020

Table 115: Number and Percentage of Subjects with Adverse Events by ALDH2 Status – Safety Subjects

| MedDRA System Organ Class/ | <b>ALDH2 Deficient</b> | <b>ALDH2 Non-deficient</b> | |
|---|---|---|---|
| Preferred Term | (N=xx) | (N=xx) | p-value |
| - Any Adverse Events - | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| SOC | | | |
| - Overall - | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Preferred term 1 | xx (xx.x%) | xx (xx.x%) | |
| Preferred term 2 | xx (xx.x%) | xx (xx.x%) | |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

p-value from chi-square test (c), unless a row has expected fewer than 5 in a cell then Fisher's exact test (f)

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 116: Number and Percentage of Subjects with Adverse Events by Treatment Arm - ALDH2 Deficient Subjects
Same analysis as Table 113

# Table 117: Number and Percentage of Subjects with Adverse Events by Treatment Arm p-values - ALDH2 Deficient Subjects

Same analysis as Table 114

# Table 118: Number and Percentage of Subjects with Adverse Events by Treatment Arm - ALDH2 Non-Deficient Subjects Same analysis as Table 113

Table 119: Number and Percentage of Subjects with Adverse Events by Treatment Arm p-values - ALDH2 Non-Deficient Subjects

Same analysis as Table 114

Table 120: Number and Percentage of Subjects Taking Drugs with Potential for Interaction

| Placebo | ANS 6637-200 mg | ANS-6637 600 mg | |
|------------|-----------------|-----------------|---------|
| (N=xx) | (N=xx) | (N=xx) | p-value |
| xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |

p-value from chi-square test

Programmer note: add a footnote of the drugs that are included

**Table 121:** Elicited Adverse Event Questions – Safety Subjects

| | Placebo | ANS-6637-200mg | ANS-6637 600 mg | Total |
|---|---|---|---|---|
| | (N=xx) <sup>1</sup> | (N=xx) | (N=xx) | (N=xx) |
| Changes in Appetite | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Heat Sensation (flushing or feeling hot) while drinking alcohol | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Heart Rate or Palpatations while drinking alcohol | xx (xx%) | xx (xx%) | xx (xx%) | xx (xx%) |

<sup>&</sup>lt;sup>1</sup>Number and percentage of subjects reporting this elicited AE.

**Table 122:** Elicited Adverse Event Questions p-values – Safety Subjects

| | ANS-6637-200mg vs<br>Placebo | ANS-6637-600mg vs<br>Placebo | ANS-6637 200 mg vs ANS-<br>6637 600 mg |
|---|---|---|---|
| Changes in Appetite | 0.xxx | 0.xxx | 0.xxx |
| Heat Sensation (flushing or feeling hot) while drinking alcohol | 0.xxx | 0.xxx | 0.xxx |
| Heart Rate or Palpatations while drinking alcohol | 0.xxx | 0.xxx | 0.xxx |

p-value from chi-square test

**Table 123:** Number of Elicited Adverse Events – Safety Subjects

| | Placebo | ANS-6637-200mg | ANS-6637 600 mg |
|---|---|---|---|
| Changes in Appetite | xx | xx | xx |
| Heat Sensation (flushing or feeling hot) while drinking alcohol | xx | xx | XX |
| Heart Rate or Palpatations while drinking alcohol | xx | xx | xx |

Number of response, not number of subjects

Table 124: Summary of Subjects with Adverse Events by Severity and Relationship – Placebo

| | Number of Subjects (%) (N=x) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mild Moderate Severe Life-threatening All Grades | | | | | | | | ; | | | |
| SOC | MedDRA<br>PT | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| | | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 125: Summary of Subjects with Adverse Events by Severity and Relationship – ANS-6637 200 mg

| | Number of Subjects (%) (N=x) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mild Moderate Severe Life-threatening All Grades | | | | | | | | | | | |
| soc | MedDRA<br>PT | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| | | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 126: Summary of Subjects with Adverse Events by Severity and Relationship – ANS-6637 600 mg

| | Number of Subjects (%) (N=x) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | M | ild | Mod | erate | Sev | ere | Life-thr | eatening | | All Grades | ; |
| soc | MedDRA<br>PT | R | NR | R | NR | R | NR | R | NR | R | NR | R + NR |
| | | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) | xx<br>(xx.x%) |

Notes: Events are counted once per subject at the highest severity grade and closest relationship to the investigational product. R= related to investigational product (possibly, probably, definitely). NR = not related to investigational product (unrelated, unlikely).

Table 127: Number and Percentage of Subjects with Adverse Events by Maximum Severity - Safety Subjects

Mild

MedDRA SOC/ Placebo
Preferred Term (N=xx)

Life-

| A A 1 | ( 0/) | ( 0/2 | ( 0/2 | 6 0/2 |
|------------------------|------------|------------|------------|------------|
| - Any Adverse Events - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| 500 | | | | |
| SOC | | | | |
| 0 11 | 6 0(2 | ( 0() | ( 0() | ( 0() |
| - Overall - | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| | | 6 0/2 | 6 0() | 6 0/2 |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Moderate

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

#### Repeat for ANS 6637-600 mg and ANS-6637 200 mg

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

threatening

Severe

Table 128: Number and Percentage of Subjects Adverse Events by Relatedness - Safety Subjects

MedDRA SOC/ Placebo ANS 6637 - 200 mg ANS-6637 600 mg (n=xx) **Preferred Term** (n=xx)(n=xx)Related1 Not-Related<sup>2</sup> Related **Not-Related** Related **Not-Related** SOC nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%) - Overall -Preferred term 1 nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%) nn(xx.x%)Preferred term 2 nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%) nn (xx.x%)

<sup>&</sup>lt;sup>1</sup>Related are possibly, probably or definitely related to investigational product

<sup>&</sup>lt;sup>2</sup> Not Related to investigational product (not related or unlikely)

Table 129: Number and Percentage of Subjects with Treatment-Related Adverse Events by Maximum Severity- Safety Subjects

MedDRA SOC/ Placebo

Preferred Term (N=xx)

| | Mild | Moderate | Severe | Life-<br>threatening |
|---|---|---|---|---|
| SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

#### Repeat for ANS 6637-600 mg and ANS-6637 200 mg

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 130: Number and Percentage of Subjects with Adverse Events Occurring in >= 10% of Subjects in Any One Group - Safety Subjects

| MedDRA SOC/ | Placebo | ANS 6637-200 mg | ANS-6637 600 mg |
|------------------|------------|-----------------|-----------------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term. At least 5% occurring in either arm to be included in the table.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 131: Number and Percentage of Subjects with Adverse Events Occurring in >= 10% of Subjects in Any One Group p-values - Safety Subjects

| MedDRA SOC/ | | | |
|---|---|---|---|
| Preferred Term | ANS-6637-200mg<br>vs Placebo | ANS-6637-600mg<br>vs Placebo | ANS-6637 200 mg<br>vs ANS-6637 600<br>mg |
| SOC | 0.xxx | 0.xxx | 0.xxx |
| - Overall - | | | |
| Preferred term 1 | 0.xxx | 0.xxx | 0.xxx |
| Preferred term 2 | 0.xxx | 0.xxx | 0.xxx |

p-values from Fisher's exact test

Table 132: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study - Safety Subjects

| MedDRA SOC/ | Placebo | ANS 6637-200 mg | ANS-6637 600 mg |
|------------------|------------|-----------------|-----------------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.

Table 133: Number and Percentage of Subjects with Adverse Events Leading to Discontinuation of Study Medication – Safety Subjects

| MedDRA SOC/ | Placebo | ANS 6637-200 mg ANS-6637 60 | |
|---|---|---|---|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| SOC | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| - Overall - | | | |
| Preferred term 1 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Preferred term 2 | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

Notes: Percentages are based on the total number of subjects, as given in the column heading.

Multiple occurrences of a specific adverse event for a subject are counted once in the frequency for the adverse event. Likewise, multiple occurrences of adverse events within a specific preferred term for a subject are counted once in the frequency for the preferred term.

Programmer's Notes: Order System Organ Class alphabetically and preferred term alphabetically within System Organ Class.
Table 134: CIWA-AR Score  $\geq$  10 at Least Once During Treatment – Safety Subjects

| | Placebo | ANS 6637-<br>200 mg | ANS-6637<br>600 mg | | | | 95% | CI <sup>2</sup> |
|---|---|---|---|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | p-value <sup>1</sup> | Cohen's h | <b>Odds Ratio</b> | OR <sup>3</sup> Lower CI | OR Upper CI |
| CIWA-AR Score >= 10 | | | | | | | | |
| Never | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | | | | |
| At Least Once | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx | | | | |
| 200 mg vs Placebo | | | | | 0.xx | xx.xxx | XX.XXX | XX.XXX |
| 600 mg vs Placebo | | | | | 0.xx | xx.xxx | XX.XXX | XX.XXX |
| 200 mg vs 600 mg | | | | | 0.xx | xx.xxx | xx.xxx | xx.xxx |

<sup>1</sup> Chi-squared test; <sup>2</sup> CI is confidence interval; <sup>3</sup> OR is odds ratio

**Table 135:** Summary of Vital Signs and Body Weights – Safety Subjects

| Parameter | N | Mean | SD | Med | Max | Min |
|--------------------|---|------|----|-----|-----|-----|
| Vital Sign (units) | | | | | | |

| Screening | | | | | | |
|----------------------|----|------|------|------|------|------|
| Placebo | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| 200 mg | xx | XX.X | xx.x | XX.X | XX.X | XX.X |
| 600 mg | XX | XX.X | XX.X | XX.X | XX.X | XX.X |
| Week 2 | | | | | | |
| Placebo | XX | XX.X | xx.x | XX.X | xx.x | XX.X |
| 200 mg | xx | XX.X | xx.x | XX.X | xx.x | XX.X |
| 600 mg | xx | XX.X | xx.x | XX.X | xx.x | XX.X |
| Change from baseline | | | | | | |
| Placebo | xx | XX.X | xx.x | XX.X | xx.x | XX.X |
| 200 mg | xx | XX.X | xx.x | XX.X | xx.x | XX.X |
| 600 mg | xx | XX.X | xx.x | XX.X | XX.X | XX.X |
| Weeks 3,4,5,6 | | | | | | |

Programmers note: vital signs include pulse rate, systolic blood pressure, and diastolic blood pressure. Body weight (kg) will also be presented.

 Table 136:
 Summary of ECG Results - Safety Subjects

| | Placebo | ANS 6637-200 mg | ANS-6637 600 mg |
|---|---|---|---|
| Result | (N=xx) | (N=xx) | (N=xx) |
| Screening | | | |
| Normal | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Week 3 | | | |
| Normal | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Week 6 | | | |
| Normal | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Not Clinically Significant | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |
| Abnormal, Clinically Significant | nn (xx.x%) | nn (xx.x%) | nn (xx.x%) |

**Table 137:** Summary of Blood Chemistries and Thyroid Function – Safety Subjects

| | Plac | Placebo | | | | ANS-6637 200mg | | | ANS-6637 600 mg | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean (SD) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) |
| Chemistry (units) | | | | | | | | | | | | |
| Baseline Value | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Week 2 | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) |
| Change from baseline | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | XX | xx.x (xx.x) | xx.x | (xx.x-xx.x) |
| Week 3, 4, 5, 6 | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) |

Programmers note: table will include creatinine, ALT, AST, total bilirubin, alkaline phosphate, albumin, CrCl, GGT and thyroid function tests.

**Table 138:** Summary of Urinalysis Continuous Data – Safety Subjects

| | Plac | Placebo | | | | ANS | ANS-6637 200mg | | | ANS-6637 600 mg | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | Mean (SD) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) | N | Mean (SD) | Med | (Min-Max) |
| Urinalysis (units) | | | | | | | | | | | | |
| Baseline Value | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) |
| Week 4 | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) |
| Change from baseline | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) |
| Week 7 | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | xx.x | (xx.x-xx.x) | xx | xx.x (xx.x) | XX.X | (xx.x-xx.x) |

Programmers note: table will PH, specific gravity, and glucose result, .

**Table 139:** Summary of Urine Glucose and Nitrites – Safety Subjects

| | Plac | Placebo | | 7-200mg | ANS-6637 600 mg | |
|---|---|---|---|---|---|---|
| | Positive | Negative | Positive | Negative | Positive | Negative |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Glucose | | | | | | |
| Baseline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Nitrites | | | | | | |
| Baseline | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Table 140: Summary of Urine Protein, Ketones, Billirubin, Leukocyte Esterace, and Blood – Safety Subjects

| | | Placebo | | AN | S-6637 200 | mg | ANS-6637 600 mg | | |
|---|---|---|---|---|---|---|---|---|---|
| | Baseline | Week 4 | Week 7 | Baseline | Week 4 | Week 7 | Baseline | Week 4 | Week 7 |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Blood | | | | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Trace | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ketones | | | | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Trace | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1+ (small) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2+ (medium) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ (large) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protein | | | | | | | | | |
| Negative | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Trace | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4+ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Programmer Note: Billirubin and Leukocyte Esterace follow the same as Protein

Table 141: Summary of Positive Urine Drug Tests, Preganancy Test or BAC > 0.02 Any Time During the Study– Safety Subjects

| | | Number (% Positive | e) |
|------------------------|----------|--------------------|-----------------|
| Test | Placebo | ANS 6637-200 mg | ANS-6637 600 mg |
| | (N=xx) | (N=xx) | (N=xx) |
| THC | xx (xx%) | xx (xx%) | xx (xx%) |
| Cocaine | xx (xx%) | xx (xx%) | xx (xx%) |
| Opioids | xx (xx%) | xx (xx%) | xx (xx%) |
| Methamphetamine | xx (xx%) | xx (xx%) | xx (xx%) |
| Amphetamine | xx (xx%) | xx (xx%) | xx (xx%) |
| MDMA | xx (xx%) | xx (xx%) | xx (xx%) |
| Benzodiazapines | xx (xx%) | xx (xx%) | xx (xx%) |
| Buprenorphine | xx (xx%) | xx (xx%) | xx (xx%) |
| Methadone | xx (xx%) | xx (xx%) | xx (xx%) |
| Oxycodone | xx (xx%) | xx (xx%) | xx (xx%) |
| Ethylglucuronide (EtG) | xx (xx%) | xx (xx%) | xx (xx%) |
| Pregnancy | xx (xx%) | xx (xx%) | xx (xx%) |

Statistical Analysis Plan: Protocol HLAB-002, Version 1.0 Dated: 16Mar2020

| | Number (% Positive) | | |
|---|---|---|---|
| Test | Placebo | ANS 6637-200 mg | ANS-6637 600 mg |
| | (N=xx) | (N=xx) | (N=xx) |
| BAC > 0.02 | xx (xx%) | xx (xx%) | xx (xx%) |

Table 142: Frequency of Subjects with Suicidal Ideation Any Time During the Study – Safety Subjects

| Number of Sub | Number of Subjects Reporting Suicidal Ideation by C-SSRS (%) | | | | |
|---|---|---|---|---|---|
| Placebo | ANS 6637-200 mg | ANS-6637 600<br>mg | ANS-6637-<br>200mg vs<br>Placebo | ANS-6637-<br>600mg vs<br>Placebo | ANS-6637 200<br>mg vs ANS-<br>6637 600 mg |
| (N=xx) | (N=xx) | (N=xx) | | | |
| xx (xx.x) | xx (xx.x) | xx (xx.x) | 0.xxx | 0.xxx | 0.xxx |

 Table 143:
 Return to Baseline ACQ-SF-R Scores – Safety Subjects

| | Number (% Positive) | | |
|------|---------------------|-----------------|-----------------|
| Test | Placebo | ANS 6637-200 mg | ANS-6637 600 mg |
| | (N=xx) | (N=xx) | (N=xx) |

| Screening | | | |
|--------------------------|----------|----------|----------|
| Increased Craving, n (%) | xx (xx%) | xx (xx%) | xx (xx%) |
| Week 2 | | | |
| Increased Craving, n (%) | xx (xx%) | xx (xx%) | xx (xx%) |

## 12.1.7. Exploratory Analyses

**Table 144:** Difference Between First and Second Alcohol Cues – mITT Subjects

| <b>Cue Question</b> | 1st Alcohol Cue | 2 <sup>nd</sup> Alcohol Cue | Difference | p-value <sup>1</sup> |
|---|---|---|---|---|
| Baseline | Mean (SD <sup>2</sup> ) | Mean (SD) | Mean (SD) | |
| Perfect | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Craving | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Drink now | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Turn down | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Average of 4 questions | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Week 2 | | | | |
| Perfect | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Craving | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Drink now | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Turn down | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |
| Average of 4 questions | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) | 0.xxx |

<sup>&</sup>lt;sup>1</sup>t-test; <sup>2</sup> SD is standard deviation

## 12.2. Listings

**Listing 1: Subject Disposition - All Subjects** 

| Subject<br>ID | Date of<br>Consent | Treatment<br>Group | mITT | Eval-<br>uable | Safety | Study<br>Completion | (Day) Date of<br>Study<br>Completion<br>or Early<br>Discontinuati<br>on | Reason for<br>Early<br>Discontinuation | Subject<br>confined<br>or incar-<br>cerated | Start Date/ End<br>Date of<br>incarceration |
|---|---|---|---|---|---|---|---|---|---|---|
| | | ANS 6637- | | | | | (xx) | | | ddmmmyyyy / |
| XXX | ddmmmyyyy | 200 mg | Yes | Yes | Yes | Yes | ddmmmyyyy | xxxxxx | Yes | ddmmmyyyy |
| | | ANS 6637-<br>600 mg | No | No | No | No | | | No | |
| | | Placebo | | | | | | | | |
| | | None | | | | | | | | |

Note: Day is relative to Study Day 0.

Listing 2. Enrollment and Randomization – All Consented Subjects

| Subject ID | Treatment Group | Date of Consent | Did the subject meet all eligibility criteria? | Randomized? | Date of Randomization | Kit Number |
|---|---|---|---|---|---|---|
| XXX | ANS 6637-200 mg | ddmmmyyyy | Yes | Yes | ddmmmyyyy | XXX |
| | ANS 6637-600 mg | | No | No | | |
| | Placebo | | | | | |

**Listing 3: Reason not Eligible – Screen Failures** 

| Subject ID | Criterion Type | Criterion |
|------------|--------------------|-----------|
| XXX | Inclusion Criteria | |
| | Exclusion Criteria | |

**Listing 4: Protocol Deviations – Safety Subjects** 

| Subject ID | Treatment Group | <b>Deviation Date</b> | Protocol Deviation | Details |
|---|---|---|---|---|
| | | | Subject Failed to Meet the | |
| XXX | ANS 6637-200 mg | ddmmmyyyy | Inclusion/Exclusion Criteria | |
| | ANS 6637-600 mg | | Source Documentation was Not Available | |
| | Placebo | | Pregnancy Test Not Performed | |
| | | | Required study data was not obtained or obtained late due to site error | |
| | | | Informed Consent Deviation | |
| | | | AE/SAE Reporting Deviation | |
| | | | Other Deviation: | xxxxxxxxxxxx |

Note: Only subjects with protocol deviation are listed.

Listing 5: Subjects Excluded from the Efficacy Analysis or Evaluable Set

| Subject<br>ID | Treatment<br>Group | Reason for Exclusion from mITT | Reason for Exclusion from Evaluable<br>Set |
|---|---|---|---|
| xxx | ANS 6637-200 mg | XXXXXX | |
| | ANS 6637-600 mg | | |
| | Placebo | | |

Note: Only subjects excluded from the efficacy analysis or evaluable set are listed.

**Listing 6: Demographics Data – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Gender | Age<br>(yrs) | Ethnicity | Race | Marital Status |
|---|---|---|---|---|---|---|
| | | | | | American Indian or Alaska | |
| XXX | ANS 6637-200 mg | Male | XX | Hispanic or Latino | Native | Married |
| | ANS 6637-600 mg | Female | | Not Hispanic or Latino | Asian | Divorced |
| | Placebo | | | Unknown | Native Hawaiian or Other<br>Pacific Islander | Living with Partner |
| | | | | | Black or African American | Widowed |
| | | | | | White | Separated |
| | | | | | Other | Never Married |
| | | | | | Unknown | Unknown |
| | | | | | | Missing |

| Subject<br>ID | Treatment<br>Group | Years of Formal<br>Education<br>(GED=12years) | Usual Employment<br>Pattern in the last 30<br>days | Subject's Annual<br>Household Income | Subject's Usual Occupation | ALDH2 Status |
|---|---|---|---|---|---|---|
| XXX | ANS 6637-<br>200 mg | xxx | Full-time, 35+ hrs/week | \$0-\$15,000 | Executive of large business or major professional | Deficient |
| | ANS 6637-<br>600 mg | | Part-time, regular hours | \$15,001-\$30,000 | Manager of medium business or minor professional | Non-deficient |
| | Placebo | | Part-time, irregular hours/daywork | \$30,001-\$45,000 | Administrator of large business, owner of small business, or semi-professional | |
| | | | Student | \$45,001-\$60,000 | Clerical or sales worker, technician | |
| | | | Military service | \$60,001-\$75,000 | Skilled worker | |
| | | | Unemployed | \$75,001-\$90,000 | Semi-skilled worker | |
| | | | Retired/Disabled | \$90,001-\$105,000 | Unskilled worker | |
| | | | Homemaker | \$105,001-\$120,000 | Unemployed | |
| | | | In controlled environment | >\$120,000 | Never worked | |
| | | | Unknown | Not Given | Not given | |
| | | | | | Other | |

**Listing 7: Baseline Drinking Characteristics – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Drinks/Day<br>(Days -1 to -<br>28) | Drinks/Day<br>(Days -1 to -14<br>Pre-<br>randomization) | Drinks/<br>Drinking Day<br>(Days -1 to -28) | Drinks/Drinking<br>Day (Days -1 to -<br>14 Pre-<br>randomization) | Weekly %<br>Heavy Drinking<br>Days<br>(Days -1 to -28) | Weekly % Heavy Drinking Days (Days -1 to -14 Pre- randomization) |
|---|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | XXX.X | XXX.X | xxxx | XXX.X | xxx.x | XXX.X |
| | ANS 6637-<br>600 mg | | | | | | |
| | Placebo | | | | | | |

| Subject<br>ID | Treatment<br>Group | Weekly %Very<br>Heavy Drinking<br>Days<br>(Days -1 to -28) | Weekly % Very<br>Heavy Drinking<br>Days<br>(Days -1 to -14<br>Pre-<br>randomization) | Weekly % Days<br>Abstinent<br>(Days -1 to -28) | Weekly % Days<br>Abstinent (Days<br>-1 to -14 Pre-<br>randomization) |
|---|---|---|---|---|---|
| | ANS 6637- | | | | |
| XXX | 200 mg | XXX.X | XXX.X | XXX.X | XXX.X |
| | ANS 6637- | | | | |
| | 600 mg | | | | |
| | Placebo | | | | |

Note: Exclude the three abstinent days during pre-randomization period.

**Listing 8: Baseline Smoking Characteristics – mITT Subjects** 

| Subject<br>ID | Treatment Group | Over the past week, how many days did you smoke cigarettes? | How many cigarettes on average per day? | Over the past week, how many days did you use nicotine products? |
|---|---|---|---|---|
| XXX | ANS 6637-200 mg | None | XXX | None |
| | ANS 6637-600 mg | 1, 2, 3, 4, 5 | | 1, 2, 3, 4, 5 |
| | Placebo | 6, 7 | | 6, 7 |
| | | Refused to answer | | Refused to answer |

**Listing 9: MINI DSM5 Disorders – Safety Subjects** 

| Subject<br>ID | Treatment Group | Visit Date | Diagnosis | Timeframe |
|---|---|---|---|---|
| XXX | ANS 6637-200 mg | ddmmmyyyy | XXXXXX | Current (2 weeks ) |
| | ANS 6637-600 mg | | | Past |
| | Placebo | | | Recurrent |

Note: Only subjects with a diagnosis of a disorder will be listed.

Listing 10: MINI DSM-5 AUD – Safety Subjects

| Subject<br>ID | Treatment<br>Group | Visit Date | # of Symptoms |
|---------------|--------------------|------------|---------------|
| xxx | ANS 6637-200<br>mg | ddmmmyyyy | XX |
| | ANS 6637-600<br>mg | | |
| | Placebo | | |

**Listing 11: Medical History – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Medical History<br>Term | Start Date | Ongoing |
|---|---|---|---|---|
| XXX | ANS 6637-200 mg | xxxxxxxxxx | ddmmmyyyy | No |
| | ANS 6637-600 mg | | | Yes |
| | Placebo | | | |

Programming note: Only identify items that were scored "yes"

**Listing 12: Drinking Goal – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Time | What goal have you chosen for yourself about drinking by the end of the study? | What might a typical week look like at the end of the study having achieved your goal? (number of drinks per day) | Motivation<br>to reach goal | Confidence to reach goal |
|---|---|---|---|---|---|---|---|
| | ANS 6637- | | | | XX | XX | XX |
| XXX | 200 mg | ddmmmyyyy | hh:mm | To stop drinking | | | |
| | ANS 6637- | | | | | | |
| | 600 mg | | | Reduce drinking but not stop | | | |
| | Placebo | | | | | | |

**Listing 13: Physical Exam – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Exam Date | Finding | Any abnormal finding during the physical exam? | Describe clinically significant findings |
|---|---|---|---|---|---|
| XXX | ANS 6637-200 mg | ddmmmyyyy | xxxxxxxxxx | Yes | XXXXXXX |
| | ANS 6637-600 mg | | | No | |
| | Placebo | | | | |

Programming Note: Only report the items that are abnormal

Listing 14: Daily and Weekly Standard Drink Units (TLFB) During Treatment – mITT Subjects

| | | | | | | | | | | Mean | Mean drinks/ | Heavy | % days |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Week | D1 | D2 | D3 | <b>D4</b> | D5 | D6 | <b>D7</b> | drinks/day | drinking day | drinking<br>days | abstinent |
| XXX | ANS 6637-<br>200 mg | 1 | XX | XX | XX | XX | XX | XX | XX | | | | |
| | ANS 6637-<br>600 mg | 2 | | | | | | | | | | | |
| | Placebo | 3, etc | | | | | | | | | | | |

**Listing 15: Brief Drinking Questionnaire – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Date of<br>Assessment | Date that the last day<br>of non-missing<br>drinking data was<br>collected by TLFB | This is a period of XX days since the last day of drinking data that was collected by TLFB | Did the subject<br>drink during<br>this period? | How many days<br>during this<br>period did the<br>subject drink? |
|---|---|---|---|---|---|---|
| | ANS 6637- | | | | | |
| XXX | 200 mg | ddmmmyyyy | ddmmmyyyy | XX | Yes | XX |
| | ANS 6637-<br>600 mg<br>Placebo | | | | No | |

| Subject<br>ID | Treatment<br>Group | Date of<br>Assessment | How many<br>alcoholic<br>drinks on a<br>typical day? | How many heavy<br>drinking days? | Maximum<br>number of drinks<br>on any one day? | How many days did<br>you drink this<br>maximum number? |
|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | ddmmmyyyy | xx | xx | XX | XX |
| | ANS 6637-<br>600 mg | | | | | |
| | Placebo | | | | | |

**Listing 16: Cue Reactivity – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit | Date of<br>Assessment | Assessment<br>Time | Cue | How strong is your craving to drink alcohol? | Having a drink would make things just perfect | If I could drink<br>alcohol now, I<br>would drink it |
|---|---|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | Screening | ddmmmyyyy | hh:mm | Water | XX | xx | XX |
| | ANS 6637-<br>600 mg | Week 2 | | | Alcohol 1 | | | |
| | Placebo | | | | Alcohol 2 | | | |

| Subject<br>ID | Treatment<br>Group | Visit | Cue | It would be hard<br>to turn down a<br>drink right now | How much did you like the beverage just given to you? | Sum of first 4 questions |
|---|---|---|---|---|---|---|
| | ANS 6637- | | | | | |
| XXX | 200 mg | Screening | Water | XX | XX | XX |
| | ANS 6637- | | | | | |
| | 600 mg | Week 2 | Alcohol 1 | | | |
| | Placebo | | Alcohol 2 | | | |

**Listing 17: Cue Session Beverage – mITT Subjects** 

| Subject<br>ID | Treatment Group | If subject smoked prior to cue session, time smoked | Typical<br>Beverage Brand | Typical<br>Beverage Type | Typical Alcohol<br>Beverage % ABV<br>(Used for Cue Session) |
|---|---|---|---|---|---|
| XXX | ANS 6637-200 mg | hh:mm | XXXXXX | xxxxxxx | xx |
| | ANS 6637-600 mg | | | | |
| | Placebo | | | | |

**Listing 18: Drinking Consequences and Craving Scores – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Week | CIWA-AR | ACQ-SF-R Pre | ACQ-SF-R Post | PACS | PROMIS Negative<br>Consequences |
|---|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | | XXX | XXX | XXX | xxx | XXX |
| | ANS 6637-<br>600 mg | | | | | | |
| | Placebo | | | | | | |

**Listing 19: Pittsburg Sleep Quality Index Scores – mITT Subjects** 

| Subject ID | Treatment Group | Week | Total score |
|------------|-----------------|-----------|-------------|
| XXX | ANS 6637-200 mg | Screening | xx |
| | ANS 6637-600 mg | Week 6 | |
| | Placebo | | |

**Listing 20: Smoking and Other Nicotine Use Data- mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Week | Visit Date | Over the past<br>week, how<br>many days did<br>you smoke<br>cigarettes? | On the days you smoked, how many cigarettes did you smoke on average? | How many days use nicotine products during the past week? |
|---|---|---|---|---|---|---|
| XXX | ANS 6637-200 mg | | ddmmmyyyy | х | xx | X |
| | ANS 6637-600 mg | | | | | |
| | Placebo | | | | | |

**Listing 21: MINI AUD- Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | | | | | | Item | | | | | | # of Symptoms |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | |
| XXX | ANS 6637-<br>200 mg | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | Y | |
| | ANS 6637-<br>600 mg | N | N | N | N | N | N | N | N | N | N | N | |
| | Placebo | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | |

| Item # | List of Items |
|---|---|
| 1 | a. During the times when you drank alcohol, did you end up drinking more than you planned when you started? |
| 2 | b. Did you repeatedly want to reduce or control your alcohol use? Did you try to cut down or control your alcohol use, but failed? IF YES TO EITHER, MARK YES. |
| 3 | c. On the days that you drank, did you spend substantial time obtaining alcohol, drinking, or recovering from the effects of alcohol? |
| 4 | d. Did you crave or have a strong desire or urge to use alcohol? |
| 5 | e. Did you spend less time meeting your responsibilities at work, at school, or at home, because of your repeated drinking? |
| 6 | f. If your drinking caused problems with your family or other people, did you still keep on drinking? |
| 7 | g. Were you intoxicated more than once in any situation where you or others were physically at risk, for example, driving a car, riding a motorbike, using machinery, boating, etc.? |
| 8 | h. Did you continue to use alcohol, even though it was clear that the alcohol had caused or worsened psychological or physical problems? |
| 9 | i. Did you reduce or give up important work, social or recreational activities because of your drinking? |
| 10 | j. Did you need to drink a lot more in order to get the same effect that you got when you first started drinking or did you get much less effect with continued use of the same amount? |

K1. When you cut down on heavy or prolonged drinking did you have any of the following: [increased sweating or heart rate; hand tremor or "the shakes"; trouble sleeping; nausea or vomiting; hearing or seeing things other people could not see or hear or having sensations in your skin for no apparent reason; agitation; anxiety; seizures] (If yes to 2 or more of these, check yes for this question), OR

K2. Did you drink alcohol to reduce or avoid withdrawal symptoms or to avoid being hung over? If K1 or K2 = yes, then score as yes.

**Listing 22. Exit Interview – mITT Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Did you think you<br>were receiving<br>the study drug or<br>the placebo? | What is your desire to please people? | If you had the opportunity in the future to take the study drug again, would you continue to take it for more than 5 weeks? | Did you limit your drinking because of flushing (a heat reaction or facial redness)? |
|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | ddmmmyyyy | Placebo | More than average | Yes | Yes |
| | ANS 6637- | 3333 | | | | |
| | 600 mg | | Study Drug | Average | No | No |
| | Placebo | | Don't know | Less than average | Refuse to answer | Refuse to answer |
| | | | Refuse to answer | Refuse to answer | | |

| Subject<br>ID | Treatment<br>Group | Visit Date | Did you limit<br>your drinking<br>because of<br>nausea or other<br>effects? | Did your<br>friends or<br>family<br>notice<br>flushing? | If your friends or<br>family noticed<br>flushing, did this<br>change your<br>drinking? | Did you ever<br>miss a dose of<br>medication to<br>avoid these<br>effects? | Did you use any<br>other services<br>during the study<br>to help you<br>reduce drinking? |
|---|---|---|---|---|---|---|---|
| XXX | ANS 6637-<br>200 mg | ddmmmyyyy | Yes | Yes | Yes | Yes | Yes |
| AAA | 9 | aamminyyyy | 103 | 103 | 103 | 163 | 103 |
| | ANS 6637-<br>600 mg | | No | No | No | No | No |
| | ooo mg | | 110 | - | 110 | 110 | 110 |
| | Placebo | | Refuse to answer | Refuse to<br>answer | Refuse to answer | Refuse to answer | Refuse to answer |

Listing 23: Drug Exposure from AiCure- mITT Subjects

| | Tablets Taken | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Study<br>Week | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Total<br>Taken | Total<br>Expected |
| XXX | ANS 6637-<br>200 mg | 1, 2, 3, 4,<br>5 | X | X | Х | X | X | Х | X | XX | XX |
| | ANS 6637-<br>600 mg | | | | | | | | | | |
| | Placebo | | | | | | | | | | |

**Listing 24: Drug Accountability – Safety Subjects** 

| Subject ID | Treatment Group | Bottle # | Date 1st Dispensed | Date Returned | # Tablets Returned |
|---|---|---|---|---|---|
| XXX | ANS 6637-200 mg | 1, 2, 3 | ddmmmyyyy | ddmmmyyyy | xx |
| | ANS 6637-600 mg | | | | |
| | Placebo | | | | |

**Listing 25: Take Control – mITT Subjects** 

| | | | Dates Modules Viewed | | | | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment Group | 1 | 2 | 3 | 4 | 5 | 6 | 7 |
| XXX | ANS 6637-200 mg | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy | ddmmmyyyy |
| | ANS 6637-600 mg | | | | | | | |
| | Placebo | | | | | | | |

**Listing 26: Adverse Events – Safety Subjects** 

Adverse Event (Verbatim) S: SOC

| Subject<br>ID | Treatment<br>Group | P: PT<br>Term | Start Date/<br>Day | Stop Date/<br>Day | Duration<br>in Days | Severity | Relation<br>-ship | Actions<br>Taken | Outcome | Seri<br>ous |
|---|---|---|---|---|---|---|---|---|---|---|
| | ANS 6637- | | ddmmmyyyy/ | ddmmmyyyy/ | | | | | | |
| XXX | 200 mg | Verbatim | XX | XX | | 1 | 1 | 1 | 1 | Yes |
| | ANS 6637- | | | | | | | | | |
| | 600 mg | S: xxxx | XX | XX | | 2 | 2 | 2 | 2 | No |
| | Placebo | P: xxxx | | | | 3 | 3 | 3 | 3 | |
| | | | | | | 4 | 4 | 4 | 4 | |
| | | | | | | | 5 | 5 | 5 | |
| | | | | | | | | 6 | | |

Notes: Day is relative to Study Day 0.

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening. Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Action Taken Due to AE: 1=None; 2=Treated with Drugs; 3=Non-drug treatment; 4=ER/Outpatient visit; 5=Hospitalization; 6=Referral for treatment

Outcome: 1=Resolved; 2=Recovered with sequelae; 3=Ongoing; 4=Required treatment; 5=Unknown

Programmer's Note: If "Were any AEs reported?" checkbox=No, then display "None Reported" in the Adverse Event column and SOC/PT column. If an AE started and stopped the same day, the duration is 1 day.

Listing 27: Adverse Events – Subjects Taking CYP3A Substrate

Adverse Event (Verbatim) S: SOC

| Subject<br>ID | Treatment<br>Group | P: PT<br>Term | Start Date/<br>Day | Stop Date/<br>Day | Duration in Days | Severity | Relation-<br>ship | Actions<br>Taken | Outcome | Serious |
|---|---|---|---|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | Verbatim | ddmmmyyyy | ddmmmyyyy | | 1 | 1 | 1 | 1 | Yes |
| | ANS 6637-<br>600 mg | S: xxxx | XX | XX | | 2 | 2 | 2 | 2 | No |
| | Placebo | P: xxxx | | | | 3 | 3 | 3 | 3 | |
| | | | | | | 4 | 4 | 4 | 4 | |
| | | | | | | | 5 | 5 | 5 | |
| | | | | | | | | 6 | | |

Notes: Day is relative to Study Day 0.

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening.

Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely

Action Taken Due to AE: 1=None; 2=Treated with Drugs; 3=Non-drug treatment; 4=ER/Outpatient visit; 5=Hospitalization; 6=Referral for treatment

Outcome: 1=Resolved; 2=Recovered with sequelae; 3=Ongoing; 4=Required treatment; 5=Unknown

Programmer's Note: If "Were any AEs reported?" checkbox=No, then display "None Reported" in the Adverse Event column and SOC/PT column. If an AE started and stopped the same day, the duration is 1 day.

**Listing 28: Serious Adverse Events – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | SAE<br>Verbatim<br>S: SOC<br>P: PT | Start Date/<br>Day | Stop Date/<br>Day | SAE Category | SAE<br>Description | Relevant<br>tests/<br>laboratory<br>data |
|---|---|---|---|---|---|---|---|
| | ANS 6637- | W 1 | 1.1 | 1.1 | D. Je : D. d | | |
| XXX | 200 mg ANS 6637- | Verbatim | ddmmmyyyy | ddmmmyyyy | Results in Death | | XXXXXX |
| | 600 mg | S: XXX | Xx | Xx | Life-threatening | | |
| | Placebo | P: XX | | | Requires or Prolongs<br>Hospitalization | | |
| | | | | | Disability | | |
| | | | | | Congenital Anomaly/Birth<br>Defect | | |
| | | | | | Required Intervention to Prevent | | |
| | | | | | Persistant or Significant<br>Disability / Incapacity | | |
| | | | | | Other | | |
| Subject<br>ID | SAE | Date of death | Cause of death | Hospitalization<br>Date/Discharge<br>Date | Comments |
|---|---|---|---|---|---|
| XXX | Verbatim | ddmmmyyyy | XXXXXX | ddmmmyyyy | xxxxxxxxxxxxxxxxxx |
| | | | | ddmmmyyyy | |

Notes: Day is relative to Study Day 0.

Severity: 1=Mild; 2=Moderate; 3=Severe; 4=Potentially Life-threatening.
Relationship: 1= Unrelated; 2=Unlikely; 3=Possibly; 4=Probably; 5=Definitely
Outcome: 1=Recovered/Resolved; 2=Recovering/Resolving; 3=Not Recovered/Not Resolved; 4=Recovered/Resolved With Sequelae; 5=Fatal (Date of Death)

**Listing 29: Elicited Adverse Events – Safety Subjects** 

| Subject<br>ID | Treatment Group | Date | Changes in appetite | Heat sensation (flushing or feeling hot) | Increased heart rate or heart palpitations |
|---|---|---|---|---|---|
| XXX | ANS 6637-200 mg | ddmmmyyyy | Yes | Yes | Yes |
| | ANS 6637-600 mg | | No | No | No |
| | Placebo | | | | |

**Listing 30: POMS Scores – mITT Subjects** 

| Subject | Treatment | Week | Total Mood | | Depressio | Scores | | | |
|---|---|---|---|---|---|---|---|---|---|
| ID | Group | | Disturbance | Tension | n | Anger | Fatigue | Confusion | Vigor |
| XXX | ANS 6637- | | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| | 200 mg | | | | | | | | |
| | ANS 6637- | | | | | | | | |
| | 600 mg | | | | | | | | |
| | Placebo | | | | | | | | |

Listing 31. Columbia-Suicide Severity Scale – Safety Subjects

| | | | | Respons | se to Ques | tion: | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | Q1 | Q2 | Q3 | Q4 | Q5 | Q6 | Q7 | Q8 | Q9 | Q10 | Q11 | Q12 | Q13 |
| xxx | ANS 6637-<br>200 mg | ddmmmyyyy | | Yes | Yes | Yes | Yes | Yes | Yes | Type 1 | 1 | 1 | 0 | 0 | 0 | Yes |
| | ANS 6637-<br>600 mg | | | No | No | No | No | No | No | Type 2 | 2 | 2 | 1 | 1 | 1 | No |
| | Placebo | | | | | | | | | Type 3 | 3 | 3 | 2 | 2 | 2 | |
| | | | | | | | | | | Type 4 | 4 | 4 | 3 | 3 | 3 | |
| | | | | | | | | | | Type 5 | 5 | 5 | 4 | 4 | 4 | |
| | | | | | | | | | | | | | 5 | 5 | 5 | |

#### **Suicide Ideation**

- 1. Have you wished you were dead or wished you could go to sleep and not wake up?
- 2. Have you actually had any thoughts of killing yourself?
- $3. \quad \text{Have you been thinking about how you might do this?} \\$
- 4. Have you had these thoughts and had some intention of acting on them?
- $5. \quad \text{Have you started to work out or worked out the details of how to kill yourself?}$
- $6. \quad \text{Do you intend to carry out this plan?} \\$

### **Intensity of Ideation**

- 7. The following features should be rated with respect to the most severe type of ideation (i.e. 1-5 with 1 being the least severe and 5 being the most severe)
- 8. How many times have you had these thoughts?1=Less than once a week; 2=Once a week; 3=2-5 times a week; 4=Daily or almost; 5=Many times each day
- 9. When you have the thoughts, how long do they last? 1=Fleeting-few seconds or minutes; 2=Less than 1 hr-some of the time; 3=1-4 hrs/a lot of time; 4=4-8 hrs/most of day; 5=More than 8 hours/persistent or continuous

- 10. Could/can you stop thining about killing yourself or wanting to die if you want to? 1=Easily; 2=Little Difficulty; 3=Some Difficulty; 4=Lot of Difficulty; 5=Unable to control; 0=Does not attempt to control
- 11. Are there things that stop you from wanting to die or acting on thoughts of committing suicide? 1=Definite deterrents; 2=Probably Deterrents; 3=Uncertain Deterrents; 4=Unlikely Deterrents; 5=No Deterrents; 0=Does not apply
- 12. What sort of reasons did you have for thinking about wanting to die or killing yourself? Was it to end pain or stop the way you were feeling or to get attention, revenge or reaction from others 1=Completely to get attention or revenge or reaction; 2=Mostly to get attention or revenge or reaction; 3=Equally to get attention or revenge or reaction and stop pain; 4=Mostly to stop pain; 5=Completely to stop pain; 0=Does not apply

### **Suicidal Behavior**

13. Have you made a suicide attempt?

| | | | Response | to Ques | tion: | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Treatment<br>Group | Study<br>Week | Q14 | Q15 | Q16 | Q17 | Q18 | Q19 | Q20 | Q21 | Q22 | Q23 | Q24 |
| XXX | ANS 6637-<br>200 mg | | XX | Yes | Yes | xx | Yes | xx | Yes | Yes | Yes | 0 | 0 |
| | ANS 6637-<br>600 mg | | | No | No | | No | | No | No | No | 1 | 1 |
| | Placebo | | | | | | | | | | | 2 | 2 |
| | | | | | | | | | | | | 3 | |
| | | | | | | | | | | | | 4 | |
| | | | | | | | | | | | | 5 (date ddmmmyyyy) | |

- 14. Number of attempts
- 15. Has the subject engaged in non-suicidal self-injurious behavior?
- 16. Has there been a time when you started to do something to end your life but someone or something stopped you before actually did anything?
- 17. Number interrupted
- 18. Has there been a time when you stared to do something to try to end your life but you stopped yourself before you actually did anything?

- 19. Number aborted
- 20. Have you taken any step towards making a suicide attempt or preparing to kill yourself?
- 21. Suicidal behavior was present during the assessment period
- 22. Completed suicide?
- 23. Actual Lethality/Medical Damage; 0=No physical damage; 1=Minor physical damage; 2=Moderate physical Damage; 3=Moderately severe physical damage; 4=Severe physical damage; 5=Death
- 24. Potential Lethality; 0=Behavior not likely to result in injury; 1=Behavior likely to result in injury, but not death; 2=Behavior likely to result in death

Listing 32: Blood Chemistries and Thyroid Results – Safety Subjects

| Subject<br>ID | Treatment Group | Visit Date | Test Name | Result | Units | Flag | Evaluation |
|---|---|---|---|---|---|---|---|
| xxxx | ANS 6637-200 mg | ddmmmyyyy | Creatinine | x.xx | mg/dL | H (high) | WNL |
| | ANS 6637-600 mg | | Total Bilirubin | XXX | mg/dL | L (low) | Abnormal, NCS |
| | Placebo | | ALT<br>AST | | U/L | | Abnormal, CS |
| | | | | X.XX | U/L | | |
| | | | Creatinine Clearance | XXX.XX | mL/min | | |
| | | | Akaline Phosphate | XXX.X | U/L | | |
| | | | Albumin | XX.X | g/dL | | |
| | | | GGT | XX.X | U/L | | |
| | | | TSH | XX.XX | | | |
| | | | Thyroxine | XX.XX | | | |
| | | Free Thyroxine | | XX.XX | | | |
| | | | Triiodothyronine | XX.XX | | | |

**Listing 33: Hematology – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Test Name | Result | Units |
|---|---|---|---|---|---|
| xxxx | ANS 6637-<br>200 mg | ddmmmyyyy | Hematocrit | xxx.xx | % |
| | ANS 6637-<br>600 mg | | Hemoglobin | xxx | g/dL |
| | Placebo | | RBC | XX.X | mil/uL |
| | | | WBC | X.XX | thous/uL |
| | | | Platelets | xxx.xx | thous/uL |
| | | | Neutrophils | XXX.X | % |
| | | | Monocytes | XX.X | % |
| | | | Eosinophils | XX.X | % |
| | | | Basophils | XX.X | % |

**Listing 34: Urinalysis – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | pН | Specific<br>Gravity | Glucose | Glucose<br>Result<br>(mg/dL) | Protein | Ketones | Blood | Nitrites | Bilirubin | Leukocyte<br>Esterase |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | ddmmmyyyy | Screen | XX.X | x.xxx | Negative | xxxx | Negative | Negative | Negative | Negative | Negative | Negative |
| | ANS 6637-<br>600 mg | | X | | | Positive | | Trace | Trace | Trace | Positive | Trace | Trace |
| | Placebo | | | | | | | 1+ | 1+ | 1+ | | 1+ | 1+ |
| | | | | | | | | 2+ | 2+ | 2+ | | 2+ | 2+ |
| | | | | | | | | 3+ | 3+ | 3+ | | 3+ | 3+ |
| | | | | | | | | 4+ | 4+ | 4+ | | 4+ | 4+ |

**Listing 35: Urinalysis Microscopy**<sup>1</sup> – **Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Test Name | Result (cells/HPF) |
|---|---|---|---|---|
| xxxx | ANS 6637-200 mg | ddmmmyyyy | Microscopic RBC | xx |
| | ANS 6637-600 mg | | Microscopic WBC | XX |
| | Placebo | | Epithelial Cells | XX |
| | | | Hyaline Casts | xx |

<sup>&</sup>lt;sup>1</sup>Only subjects that had microscopy

Listing 36: Pregnancy Test/Birth Control Data – Safety Subjects

| Subject<br>ID | Treatment Group | Gender | Pregnancy Test Performed? | Pregnancy Test /<br>Visit Date | Pregnancy Result | Methods of birth control |
|---|---|---|---|---|---|---|
| XXX | ANS 6637-200 mg | Male | Not Done | ddmmmyyyy | Negative | Oral Contraceptive |
| | ANS 6637-600 mg | Female | Yes | | Positive | Contraceptive Sponge |
| | Placebo | | | | | Contraceptive Skin Patch |
| | | | | | | Double Barrier |
| | | | | | | Intrauterine |
| | | | | | | Etonogestrel implant |
| | | | | | | Medroxyprogesterone |
| | | | | | | Complete Abstinence |
| | | | | | | Hormonal Viginal contraceptive Ring |
| | | | | | | Surgically Sterile |
| | | | | | | Postemopausal |
| | | | | | | Partner surgically Sterile |
| | | | | | | Other: xxxxxxxxxxxxxxx |

Programming note: Only indicate birth control methods that were indicated as Yes

**Listing 37: Blood Alcohol Concentration – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Visit Date | Study<br>Week | BAC<br>Performed | Time of<br>BAC | BAC % |
|---|---|---|---|---|---|---|
| xxx | ANS 6637-200<br>mg | ddmmmyyyy | х | Done | hh:mm | x.xxx |
| | ANS 6637-600<br>mg | | | Not Done | | |
| | Placebo | | | | | |

**Listing 38. Urine Drug Screen – Safety Subjects** 

| Subject ID | Treatment<br>Group | Visit Date | Study<br>Week | AMP <sup>1</sup> | Benzos <sup>2</sup> | Coc <sup>3</sup> | Bup <sup>4</sup> | Meth <sup>5</sup> | Methadone | Opioids | ТНС | Barb <sup>6</sup> | MDMA | EtG <sup>7</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | ddmmmyyyy | Screen | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg | Neg |
| | ANS 6637-<br>600 mg | | X | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos | Pos |
| | Placebo | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup>AMP = Amphetamine; <sup>2</sup>Benzos = Benzodiazapines; <sup>3</sup> Coc = Cocaine; <sup>4</sup> Bup = Buprenorphine; <sup>5</sup> Methamphetamine; <sup>6</sup>Barb = Barbituates;

<sup>&</sup>lt;sup>7</sup> EtG = Ethyl Glucuronide; Note: Neg=negative; Pos=positive

Listing 39: Vital Signs and Body Weights-Safety Subjects

| Subject ID | Treatment<br>Group | Visit Date | Study<br>Week | Weight (Kg) | Heart Rate<br>(beats/min) | Systolic Pressure<br>(mmHg) | Diastolic Pressure<br>(mmHg) |
|---|---|---|---|---|---|---|---|
| | ANS 6637-200 | | | | | | |
| XXX | mg | ddmmmyyyy | Screening | XXX | xxx | XXX | XXX |
| | ANS 6637-600<br>mg | | x | | | | |
| | Placebo | | | | | | |

**Listing 40. ECG – Safety Subjects** 

| Subject ID | Treatment Group | Visit Date | Study<br>Week | Result | If abnormal, specify finding |
|---|---|---|---|---|---|
| xxx | ANS 6637-200<br>mg | ddmmmyyyy | Screen 1 | Normal | xxxxxxxxx |
| | ANS 6637-600<br>mg | | x | Abnormal, NCS | |
| | Placebo | | | Abnormal, CS | |

Listing 41. Prior and Concomitant Medications – Safety Subjects

| Subject<br>ID | Treatment<br>Group | Special<br>Med<br>Class | Verbatin Med | Indication | Route | Frequency | Dose | Start Date/<br>Stop Date | Study Day | Continuing? |
|---|---|---|---|---|---|---|---|---|---|---|
| | ANS<br>6637-200 | | | xxxxxx | | xxxxxx | | ddmmmyyyy | xxx | |
| xxx | mg<br>ANS<br>6637-600<br>mg | Yes | XXX | | XXXXXX | | xxxxxx | | | Yes |
| | Placebo | No | xxx | | | | | | | No |

A special med is one that has potential for drug-drug interactions. Classes of these medications include proton pump inhibitors, histamine-2 antagonists,. OATP1B1 and OATP1B3 transporters, OAT1 and OAT3 transporters, MATE1, MATE-2K, and OCT2 transporters, P-gp transporter tnhibitors, and BCRP transporters.

**Listing 42: Blood for Drug Concentrations – Safety Subjects** 

| Subject<br>ID | Treatment<br>Group | Sample<br>Collected? | PK Sampling<br>Date | PK Sampling Time | Sampling Problems? | GS-548351<br>Plasma Level<br>(ng/mL) | Comments |
|---|---|---|---|---|---|---|---|
| xxx | ANS 6637-<br>200 mg | Yes | ddmmmyyyy | hh:mm | Yes | | xxxxxx |
| | ANS 6637-<br>600 mg | No | | | No | | |
| | Placebo | | | | | | |

**Listing 43: Comments – Safety Subjects** 

| Subject ID | Treatment Group | Comments |
|------------|-----------------|--------------|
| xxx | ANS 6637-200 mg | XXXXXXXXXXXX |
| | ANS 6637-600 mg | |
| | Placebo | |

# 12.3. Figures

### Figure 1: Percentage of Subjects No Heavy Drinking Days Weeks 2-5

Programmer note: Use percent on y-axis, bar graph of PSNHDD add Cohen's h, \* a significant p-value, put values on graph

### Figure 2: Percentage of Subjects Abstinent Weeks 2-5

Programmer note: bar graph of PSA add Cohen's h, \* a significant p-value, put values on graph

## Figure 3: Weekly Percentage of Subjects No Heavy Drinking Days (mITT)

Programmer note: graph of estimates out to 5 weeks. Include 95% confidence intervals for each estimate and \* on statistically significant differences between treatment groups.

- Figure 4: Weekly Percentage of Subjects Abstinent (mITT)
- Figure 5: Weekly Percentage WHO 1-Level Decrease in Alcohol Consumption (mITT)
- Figure 6: Weekly Percentage WHO 2-Level Decrease in Alcohol Consumption No Imputation (mITT)
- Figure 7: Percentage Days Abstinent per Week Least Squares Means (mITT)
- Figure 8: Percent Heavy Drinking Days per Week Lease Squares Means –(mITT)
- Figure 9: Mean Drinks per Week Lease Squares Means (mITT)
- Figure 10: Mean Drinks per Drinking Day by Week Least Squares Means (mITT)
- Figure 11: Weekly Number of Cigarettes Smoked in Smokers Over Entire Treatment Period Least Squares Means (mITT)
- Figure 12: Clinical Chemistry, Urinalysis, and Hematology Values Over Time